CLINICAL TRIAL: NCT00263328
Title: A Multicenter, Phase 2, Open-label, Controlled, Extension Study For Stage 1 Subjects Of Study A3921009 To Evaluate The Long-term Safety And Efficacy Of Cp-690,550 Versus Tacrolimus, When Co-administered With Mycophenolate Mofetil In Renal Allograft Recipients
Brief Title: Extension Study Of Stage 1 Subjects Of Study A3921009 For The Prevention Of Acute Rejection In Kidney Transplant Patient
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3921021
Record Dates: First submitted 2005-12-06; First posted 2005-12-08 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Kidney Transplantation
Keywords: immunosuppression; JAK3 inhibitor; kidney transplant; tofacitinib; Xeljanz; CP-690; 550; tacromilus; mycophenolate mofetil
MeSH Terms: interventions — Tacrolimus; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment group 1 (Active Comparator): Standard of care
  Interventions: Drug: Tacrolimus
- Treatment group 2 (Experimental): Treatment group 2 also receives mycophenolate mofetil
  Interventions: Drug: CP-690,550
- Treatment group 3 (Experimental): Treatment group 3 does not receive mycophenolate mofetil
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Tacrolimus — Standard of care
  Arms: Treatment group 1
Drug: CP-690,550 — CP-690,550 5 mg BID
  Arms: Treatment group 2
Drug: CP-690,550 — CP-690,550 10 mg BID
  Arms: Treatment group 3

SUMMARY:
A new immunosuppressive drug, based on the inhibition of an important enzyme in the immune system called JAK3, is being developed by Pfizer to prevent transplant rejection. In study A3921009, kidney transplant patients were given a JAK inhibitor or tacrolimus for 6 months posttransplant. Patients who completed study A3921009 were offered the opportunity to participate in study A3921021 which will extend the evaluation of safety and efficacy of CP-690,550 versus tacrolimus through 8 years posttransplant. In treatment group 1 (control arm), subjects will continue to receive tacrolimus. In treatment groups 2 and 3, subjects will continue to receive CP-690,550. Per Amendment 4, the tacrolimus comparator arm will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in Stage 1 of Study A3921009 and have completed 6-months of treatment with trial medications (CP-690,550 or tacrolimus)
* Recipient of a first-time kidney transplant

Exclusion Criteria:

* Subject with any untreated condition that may affect drug absorption (eg, gastrectomy or clinically significant diabetic gastroenteropathy).
* Subjects who are on the waiting list for a second kidney transplant or any non-renal organ transplants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-12; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (27):
  - Multi Organ Transplant Center, Los Angeles, California
  - St. Vincent Medical Center, Los Angeles, California
  - Transplant Research Institute, Los Angeles, California
  - Stanford School of Medicine, Palo Alto, California
  - Balboa Institute of Transplantation, San Diego, California
  - California Institute of Renal Research, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, Kidney Transplant Unit, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Sciences Center Renal Clinical Trials Office, Aurora, Colorado
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University-Feinberg School of Medicine, Division of Organ Transplantation, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Jack J Dreyfus Clinic, New York, New York
  - Recanati/Miller Transplantation Institute, New York, New York
  - New York Presbyterian Hospital / Weill Cornell Medical Center, New York, New York
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Legacy Transplant Services, Portland, Oregon
  - Northwest Renal Clinic, Portland, Oregon
  - Dallas Transplant Institute, Dallas, Texas
  - Annette C & Harold C Simmons Transplant Institute, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Busque S, Leventhal J, Brennan DC, Steinberg S, Klintmalm G, Shah T, Mulgaonkar S, Bromberg JS, Vincenti F, Hariharan S, Slakey D, Peddi VR, Fisher RA, Lawendy N, Wang C, Chan G. Calcineurin-inhibitor-free immunosuppression based on the JAK inhibitor CP-690,550: a pilot study in de novo kidney allograft recipients. Am J Transplant. 2009 Aug;9(8):1936-45. doi: 10.1111/j.1600-6143.2009.02720.x. PMID 19660021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921021&StudyName=Extension%20Study%20Of%20Stage%201%20Subjects%20Of%20Study%20A3921009%20For%20The%20Prevention%20Of%20Acute%20Rejection%20In%20Kidney%20Transplant%20Patient

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus: Participants received tacrolimus BID, administered according to standard institutional practice up to 72 months. Tacrolimus dosage was adjusted to achieve pre-determined target predose (trough) tacrolimus levels in whole blood (5-12 ng/mL through 12 months post-transplant, 3-10 ng/mL thereafter). In addition, African-American participants may have received MMF, up to 3 gm per day through Month 6 post-transplant. Participants also received corticosteroids (prednisone ≤5 mg daily [or equivalent] through at least 12 months posttransplant. Thereafter, steroids may have been discontinued at the investigator's discretion.
- Tofacitinib 15-10-5 mg BID: Participants receiving tofacitinib 15 mg, tablets, PO, BID at study entry (rollover from Parent Study A3921009) reduced the dose of tofacitinib to 10 mg BID on entry into Study A3921021. Within the window of Months 12-24 post-transplant, tofacitinib dosage was then tapered from 10 mg BID to 5 mg BID over 4 weeks (5 mg in the morning and 10 mg in the evening for 4 weeks, then 5 mg BID thereafter) and the participant remained on 5 mg BID throughout the duration of the study, for a maximum of 90 months. In addition, African-American participants may have received MMF, up to 3 gm per day through Month 6 post-transplant. Participants also received corticosteroids (prednisone ≤5 mg daily [or equivalent] through at least 12 months post-transplant. Thereafter, steroids may have been discontinued at the investigator's discretion.
- Tofacitinib 30-15-10 mg BID: Participants receiving tofacitinib 30 mg, tablets, PO, BID at study entry (rollover from Parent Study A3921009) tapered tofacitinib dosage from 30 mg BID to 15 mg BID over 4 weeks on entry into Study A3921021 (25 mg BID for 2 weeks, 20 mg BID for 2 weeks, then 15 mg BID thereafter). Within the window of Months 12-24 post-transplant, tofacitinib dosage was tapered from 15 mg BID to 10 mg BID and participants remained on 10 mg BID throughout the duration of the study, for a maximum of 90 months. Participants also received corticosteroids (prednisone ≤5 mg daily [or equivalent] through at least 12 months post-transplant. Thereafter, steroids may have been discontinued at the investigator's discretion.
Period: Overall Study
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Started | 18 | 14 | 13
Completed | 10 | 12 | 6
Not Completed | 8 | 2 | 7
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1
Not completed — Other | 3 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study medication in the study.
Groups:
- Tofacitinib: Participants received tacrolimus BID, administered according to standard institutional practice. Tacrolimus dosage was adjusted to achieve pre-determined target predose (trough) tacrolimus levels in whole blood (5-12 ng/mL through 12 months post-transplant, 3-10 ng/mL thereafter). In addition, African-American participants may have received MMF, up to 3 gm per day through Month 6 post-transplant. Participants also received corticosteroids (prednisone ≤5 mg daily [or equivalent] through at least 12 months post-transplant. Thereafter, steroids may have been discontinued at the investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID | Total
Number analyzed (Participants) | 18 | 14 | 13 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.6 (9.3) | 48.1 (7.9) | 44.5 (12.2) | 43.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 3 | 17
  Male | 11 | 7 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Calculated Glomerular Filtration Rate (GFR) Using the Modification of Diet in Renal Disease (MDRD) Equation
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using MDRD equation. GFR by MDRD equation = 170 * (serum creatinine [in milligrams per deciliter (mg/dL)])^(-0.999) * (age in years)^(-0.176) * (0.762 if female) * (1.18 if black) * (blood urea nitrogen [BUN] concentration [mg/dL])^(-0.170) * (serum albumin concentration [in grams per dL (g/dL)])^(0.318). A normal GFR is >90 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2), although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min/1.73 m^2 indicated kidney failure.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Groups:
- Tacrolimus: Participants received tacrolimus BID, administered according to standard institutional practice up to 72 months. Tacrolimus dosage was adjusted to achieve pre-determined target predose (trough) tacrolimus levels in whole blood (5-12 ng/mL through 12 months post-transplant, 3-10 ng/mL thereafter). In addition, African-American participants may have received MMF, up to 3 gm per day through Month 6 post-transplant. Participants also received corticosteroids (prednisone ≤5 mg daily [or equivalent] through at least 12 months post-transplant. Thereafter, steroids may have been discontinued at the investigator's discretion.
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mL/min/1.73 m^2
  Month 9 (n=18,14,12) | 67.06 (19.79) | 65.99 (12.46) | 67.05 (13.63)
  Month 12 (n=16,14,12) | 64.97 (25.10) | 65.16 (11.90) | 63.50 (12.01)
  Month 15 (n=16,14,12) | 66.22 (15.10) | 67.86 (9.33) | 65.71 (9.44)
  Month 18 (n=18,14,12) | 72.81 (23.09) | 66.91 (12.19) | 64.71 (12.10)
  Month 24 (n=17,14,12) | 77.05 (28.23) | 68.45 (10.47) | 66.29 (8.72)
  Month 30 (n=14,14,10) | 79.89 (29.56) | 71.55 (7.33) | 64.04 (10.24)
  Month 36 (n=15,14,9) | 79.87 (30.20) | 70.44 (13.65) | 61.72 (15.84)
  Month 42 (n=15,14,9) | 77.95 (29.77) | 70.77 (16.05) | 65.25 (8.71)
  Month 48 (n=15,14,10) | 76.23 (30.34) | 70.36 (14.36) | 65.50 (10.19)
  Month 54 (n=14,14,10) | 78.10 (32.27) | 69.98 (15.18) | 61.99 (9.54)
  Month 60 (n=13,13,10) | 82.86 (33.72) | 70.10 (18.01) | 67.30 (9.37)
  Month 66 (n=12,14,10) | 89.80 (36.51) | 69.69 (18.23) | 64.98 (15.95)
  Month 72 (n=9,13,8) | 76.61 (20.99) | 67.89 (11.61) | 61.96 (8.15)
  Month 78 (n=0,13,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 69.95 (14.40) | 68.64 (6.15)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 69.24 (13.80) | 68.77 (4.90)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 65.28 (14.19) | 69.46 (6.23)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 64.94 (14.01) | 70.33 (14.22)
  Follow-up (n=6,12,8) | 42.29 (19.87) | 63.25 (14.07) | 60.41 (24.43)

2. Primary Outcome: Serum Creatinine Levels
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mg/dL
  Month 9 (n=18,14,12) | 1.26 (0.30) | 1.19 (0.26) | 1.28 (0.31)
  Month 12 (n=16,14,12) | 1.34 (0.30) | 1.21 (0.30) | 1.33 (0.32)
  Month 15 (n=16,14,12) | 1.24 (0.32) | 1.13 (0.20) | 1.28 (0.29)
  Month 18 (n=18,14,12) | 1.18 (0.30) | 1.15 (0.23) | 1.29 (0.29)
  Month 24 (n=17,14,12) | 1.15 (0.29) | 1.11 (0.18) | 1.23 (0.22)
  Month 30 (n=14,14,10) | 1.14 (0.36) | 1.06 (0.16) | 1.24 (0.22)
  Month 36 (n=15,14,9) | 1.18 (0.43) | 1.08 (0.22) | 1.33 (0.30)
  Month 42 (n=15,14,9) | 1.19 (0.42) | 1.09 (0.27) | 1.17 (0.12)
  Month 48 (n=15,14,10) | 1.23 (0.47) | 1.08 (0.27) | 1.20 (0.11)
  Month 54 (n=14,14,10) | 1.38 (1.04) | 1.10 (0.26) | 1.25 (0.14)
  Month 60 (n=13,13,10) | 1.17 (0.40) | 1.12 (0.35) | 1.16 (0.13)
  Month 66 (n=12,14,10) | 1.12 (0.50) | 1.14 (0.33) | 1.24 (0.27)
  Month 72 (n=9,13,8) | 1.12 (0.26) | 1.09 (0.21) | 1.29 (0.21)
  Month 78 (n=0,13,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.09 (0.21) | 1.16 (0.14)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.10 (0.21) | 1.15 (0.15)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.16 (0.25) | 1.16 (0.19)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.15 (0.25) | 1.10 (0.14)
  Follow-Up (n=6,12,8) | 2.35 (2.11) | 1.16 (0.27) | 1.50 (0.84)

3. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Clinically Significant Infections by Visit
Description: Kaplan-Meier analysis of percentage of participants with clinically significant infections by time to first clinically significant infection within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 16 | 14 | 12
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=16,14,12) | 11.11 | 0.00 | 7.69
  Month 3 (n=16,13,7) | 11.11 | 7.14 | 46.15
  Month 6 (n=14,12,4) | 22.22 | 14.29 | 69.23
  Month 9 (n=13,11,4) | 27.78 | 21.43 | 69.23
  Month 12 (n=12,9,4) | 33.33 | 35.71 | 69.23
  Month 15 (n=11,8,3) | 38.89 | 42.86 | 76.92
  Month 18 (n=10,8,3) | 38.89 | 42.86 | 76.92
  Month 24 (n=10,8,3) | 38.89 | 42.86 | 76.92
  Month 30 (n=9,8,3) | 38.89 | 42.86 | 76.92
  Month 36 (n=8,8,3) | 45.68 | 42.86 | 76.92
  Month 42 (n=8,8,2) | 45.68 | 42.86 | 76.92
  Month 48 (n=7,8,2) | 45.68 | 42.86 | 76.92
  Month 54 (n=7,8,2) | 45.68 | 42.86 | 76.92
  Month 60 (n=7,8,2) | 45.68 | 42.86 | 76.92
  Month 66 (n=7,8,2) | 45.68 | 42.86 | 76.92
  Month 72 (n=4,8,2) | 45.68 | 42.86 | 76.92
  Month 84 (n=0,8,2) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 42.86 | 76.92
  Month 90 (n=0,8,2) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 42.86 | 76.92
  Month 96 (n=0,8,2) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 42.86 | 76.92

4. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With New Onset Diabetes Mellitus, Definition 1 (NODM-1) by Visit
Description: Kaplan-Meier analysis of time to NODM-1 within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. NODM-1 was defined as an event experienced by participants who were non-diabetic prior to transplantation and required treatment with oral hypoglycemic agents, anti-diabetic agents, and/or insulin for greater than or equal to (â‰¥)30 days.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; participants who had a history of diabetes at transplant were not included in the Kaplan-Meier analysis. n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 17 | 8 | 9
percentage of participants
  Month 1 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 3 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 6 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 9 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 12 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 15 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 18 (n=16,8,9) | 0.00 | 0.00 | 0.00
  Month 24 (n=15,8,9) | 6.25 | 0.00 | 0.00
  Month 30 (n=13,8,8) | 6.25 | 0.00 | 0.00
  Month 36 (n=13,8,8) | 6.25 | 0.00 | 0.00
  Month 42 (n=13,8,8) | 6.25 | 0.00 | 0.00
  Month 48 (n=12,8,8) | 6.25 | 0.00 | 0.00
  Month 54 (n=12,8,8) | 6.25 | 0.00 | 0.00
  Month 60 (n=11,8,8) | 6.25 | 0.00 | 0.00
  Month 66 (n=11,8,7) | 6.25 | 0.00 | 0.00
  Month 72 (n=6,8,7) | 6.25 | 0.00 | 0.00
  Month 78 (n=0,8,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 0.00
  Month 84 (n=0,8,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 0.00
  Month 90 (n=0,8,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 0.00
  Month 96 (n=0,8,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 0.00

5. Primary Outcome: Percentage of Participants With Hypercholesterolemia
Description: Hypercholesterolemia was defined as cholesterol levels >240 mg/dL or 6.2 mmol/L.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 9 (n=18,14,13) | 11.1 | 35.7 | 15.4
  Month 12 (n=18,14,12) | 5.6 | 28.6 | 8.3
  Month 15 (n=18,14,12) | 5.6 | 35.7 | 0
  Month 18 (n=18,14,12) | 5.6 | 7.1 | 8.3
  Month 24 (n=17,14,12) | 11.8 | 7.1 | 16.7
  Month 30 (n=15,14,11) | 6.7 | 7.1 | 9.1
  Month 36 (n=15,14,11) | 6.7 | 0 | 9.1
  Month 42 (n=15,14,10) | 6.7 | 21.4 | 0
  Month 48 (n=15,14,10) | 20.0 | 7.1 | 10.0
  Month 54 (n=14,14,10) | 14.3 | 21.4 | 10.0
  Month 60 (n=13,14,10) | 7.7 | 0 | 20.0
  Month 66 (n=12,14,10) | 16.7 | 14.3 | 0
  Month 72 (n=9,13,8) | 11.1 | 15.4 | 12.5
  Month 78 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.7 | 12.5
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.7 | 0
  Month 90 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 8.3 | 0
  Month 96 (n=0,11,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 9.1 | 0
  Follow-Up (n=7,14,11) | 14.3 | 7.1 | 9.1

6. Primary Outcome: Percentage of Participants With Hypertriglyceridemia by Visit
Description: Hypertriglyceridemia was defined as triglyceride levels of >200 mg/dL or 2.3 mmol/L.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 9 (n=18,14,13) | 11.1 | 50.0 | 38.5
  Month 12 (n=18,14,12) | 5.6 | 42.9 | 33.3
  Month 15 (n=18,14,12) | 5.6 | 42.9 | 41.7
  Month 18 (n=18,14,12) | 5.6 | 35.7 | 33.3
  Month 24 (n=17,14,12) | 17.6 | 21.4 | 33.3
  Month 30 (n=15,14,11) | 13.3 | 28.6 | 36.4
  Month 36 (n=15,14,11) | 20.0 | 14.3 | 27.3
  Month 42 (n=15,14,10) | 20.0 | 35.7 | 20.0
  Month 48 (n=15,14,10) | 20.0 | 35.7 | 30.0
  Month 54 (n=14,14,10) | 7.1 | 35.7 | 40.0
  Month 60 (n=13,14,10) | 15.4 | 0 | 30.0
  Month 66 (n=12,14,10) | 16.7 | 14.3 | 20.0
  Month 72 (n=9,13,8) | 11.1 | 23.1 | 50.0
  Month 78 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.7 | 25.0
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.7 | 37.5
  Month 90 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 8.3 | 50.0
  Month 96 (n=0,11,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 18.2 | 33.3
  Follow-Up (n=7,14,11) | 14.3 | 14.3 | 27.3

7. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With First Biopsy Proven Acute Rejection (BPAR) by Visit
Description: Kaplan-Meier analysis of percentage of participants with first BPAR by time to first BPAR within 96 months post-transplant. BPAR was defined as acute/active cellular rejection (Category 4 of the Banff Classification), based on the assessment of the renal allograft biopsy by a central, blinded pathologist. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=17,14,13) | 5.56 | 0.00 | 0.00
  Month 3 (n=17,14,11) | 5.56 | 0.00 | 15.38
  Month 6 (n=17,14,11) | 5.56 | 0.00 | 15.38
  Month 9 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 12 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 15 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 18 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 24 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 30 (n=14,14,10) | 11.11 | 0.00 | 15.38
  Month 36 (n=14,14,10) | 11.11 | 0.00 | 15.38
  Month 42 (n=14,14,9) | 11.11 | 0.00 | 15.38
  Month 48 (n=13,14,9) | 11.11 | 0.00 | 15.38
  Month 54 (n=13,14,9) | 11.11 | 0.00 | 15.38
  Month 60 (n=12,14,9) | 11.11 | 0.00 | 15.38
  Month 66 (n=12,14,8) | 11.11 | 0.00 | 15.38
  Month 72 (n=5,14,7) | 11.11 | 0.00 | 15.38
  Month 78 (n=0,14,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38
  Month 84 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38
  Month 90 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38

8. Primary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Treatment Failure by Visit
Description: Kaplan-Meier analysis of percentage of participants with treatment failure by time to treatment failure within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. Treatment failure was defined as the first occurrence of BPAR, death, graft loss or premature discontinuation of trial medication for any reason.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of study medication. n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=17,14,13) | 5.56 | 0.00 | 0.00
  Month 3 (n=17,14,11) | 5.56 | 0.00 | 15.38
  Month 6 (n=17,14,11) | 5.56 | 0.00 | 15.38
  Month 9 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 12 (n=16,14,10) | 11.11 | 0.00 | 23.08
  Month 15 (n=16,14,10) | 11.11 | 0.00 | 23.08
  Month 18 (n=16,14,10) | 11.11 | 0.00 | 23.08
  Month 24 (n=15,14,10) | 16.67 | 0.00 | 23.08
  Month 30 (n=14,14,9) | 22.22 | 0.00 | 30.77
  Month 36 (n=14,14,8) | 22.22 | 0.00 | 38.46
  Month 42 (n=14,14,8) | 22.22 | 0.00 | 38.46
  Month 48 (n=13,14,8) | 27.78 | 0.00 | 38.46
  Month 54 (n=13,14,8) | 27.78 | 0.00 | 38.46
  Month 60 (n=12,14,8) | 33.33 | 0.00 | 38.46
  Month 66 (n=11,14,8) | 38.89 | 0.00 | 38.46
  Month 72 (n=5,13,6) | 50.00 | 7.14 | 53.85
  Month 78 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 53.85
  Month 84 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 53.85
  Month 90 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 14.29 | 53.85
  Month 96 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 14.29 | 53.85

9. Secondary Outcome: Calculated GFR Using the Nankivell Equation (mL/Min)
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was estimated by creatinine clearance (CLcr; in mL/min]) using Nankivell equation. CLcr by Nankivell equation= (6.7 per serum creatinine [in millimoles per liter (mmol/L)]) plus (0.25*body weight [in kilograms (kg)]) minus (0.5*serum urea [mmol/dL, where 1 mg/dL BUN=0.36 mmol/L urea]) minus (100 per height [in meters] square) plus (35 for male/25 for female). A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mL/min
  Month 9 (n=18,14,12) | 77.98 (11.29) | 80.15 (9.74) | 81.39 (9.77)
  Month 12 (n=16,14,12) | 73.64 (15.23) | 80.02 (9.39) | 79.31 (11.71)
  Month 15 (n=16,14,12) | 80.92 (12.79) | 83.06 (6.99) | 81.18 (10.61)
  Month 18 (n=18,14,12) | 82.77 (14.14) | 81.72 (10.35) | 80.03 (10.82)
  Month 24 (n=17,14,12) | 84.93 (14.36) | 82.62 (10.15) | 81.66 (8.20)
  Month 30 (n=14,14,10) | 88.61 (16.59) | 86.35 (7.12) | 79.87 (9.74)
  Month 36 (n=15,14,9) | 89.08 (24.53) | 86.05 (12.76) | 76.38 (15.14)
  Month 42 (n=15,14,9) | 86.95 (17.96) | 86.07 (13.13) | 81.89 (7.03)
  Month 48 (n=15,14,10) | 85.59 (21.32) | 86.47 (13.32) | 82.06 (8.68)
  Month 54 (n=14,14,10) | 88.08 (27.63) | 85.35 (12.99) | 79.98 (10.36)
  Month 60 (n=13,13,10) | 93.01 (19.88) | 85.75 (15.79) | 85.36 (10.01)
  Month 66 (n=12,14,10) | 98.72 (33.70) | 84.26 (16.14) | 82.21 (17.48)
  Month 72 (n=9,13,8) | 90.60 (17.58) | 83.80 (10.92) | 81.46 (7.94)
  Month 78 (n=0,13,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 83.94 (10.95) | 87.44 (8.72)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 84.21 (12.50) | 88.53 (5.40)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 81.09 (12.75) | 88.91 (6.31)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 79.46 (12.35) | 88.20 (8.93)
  Follow-Up (n=6,12,8) | 52.35 (28.37) | 81.06 (12.76) | 76.41 (29.81)

10. Secondary Outcome: Calculated GFR Using Cockcroft-Gault Equation (mL/Min)
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using Cockcroft-Gault equation. GFR by Cockcroft-Gault equation= body weight (kg)*(140 minus age in years) divided by (72*serum creatinine [mg/dL]). For females value obtained was multiplied by 0.85. A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mL/min
  Month 9 (n=18,14,12) | 92.82 (19.95) | 86.74 (15.70) | 92.35 (10.45)
  Month 12 (n=16,14,12) | 87.05 (19.95) | 87.29 (17.83) | 90.36 (18.79)
  Month 15 (n=16,14,12) | 98.39 (22.67) | 92.69 (15.97) | 92.79 (15.98)
  Month 18 (n=18,14,12) | 98.68 (24.03) | 90.61 (16.53) | 91.31 (18.19)
  Month 24 (n=17,14,12) | 100.46 (21.65) | 89.62 (24.06) | 94.67 (16.46)
  Month 30 (n=14,14,10) | 102.29 (21.29) | 95.79 (20.38) | 88.19 (13.32)
  Month 36 (n=15,14,9) | 101.92 (33.77) | 94.67 (23.12) | 86.32 (22.76)
  Month 42 (n=15,14,9) | 102.79 (27.15) | 92.13 (19.39) | 91.96 (14.62)
  Month 48 (n=15,14,10) | 100.77 (27.37) | 92.78 (23.60) | 93.23 (19.62)
  Month 54 (n=14,14,10) | 106.65 (33.50) | 89.96 (19.19) | 91.90 (21.03)
  Month 60 (n=13,13,10) | 113.73 (31.33) | 87.89 (21.20) | 98.94 (21.29)
  Month 66 (n=12,14,10) | 118.60 (42.38) | 86.74 (20.14) | 94.80 (32.99)
  Month 72 (n=9,13,8) | 113.23 (30.03) | 86.00 (17.77) | 93.33 (18.12)
  Month 78 (n=0,13,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 85.10 (16.99) | 100.93 (20.40)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 85.54 (19.31) | 102.36 (14.46)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 80.73 (19.03) | 103.59 (16.99)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 79.02 (18.97) | 100.89 (14.55)
  Follow-Up (n=6,12,8) | 63.95 (35.17) | 82.26 (17.32) | 89.79 (40.28)

11. Secondary Outcome: Reciprocal of Serum Creatinine
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: dL/mg
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
dL/mg
  Month 9 (n=18,14,12) | 0.83 (0.17) | 0.88 (0.22) | 0.83 (0.20)
  Month 12 (n=16,14,12) | 0.78 (0.17) | 0.88 (0.22) | 0.80 (0.21)
  Month 15 (n=16,14,12) | 0.85 (0.19) | 0.91 (0.17) | 0.82 (0.20)
  Month 18 (n=18,14,12) | 0.89 (0.20) | 0.90 (0.18) | 0.81 (0.18)
  Month 24 (n=17,14,12) | 0.92 (0.22) | 0.93 (0.16) | 0.83 (0.15)
  Month 30 (n=14,14,10) | 0.95 (0.29) | 0.96 (0.14) | 0.83 (0.18)
  Month 36 (n=15,14,9) | 0.96 (0.38) | 0.96 (0.20) | 0.78 (0.14)
  Month 42 (n=15,14,9) | 0.92 (0.25) | 0.97 (0.24) | 0.87 (0.09)
  Month 48 (n=15,14,10) | 0.91 (0.27) | 0.98 (0.23) | 0.84 (0.08)
  Month 54 (n=14,14,10) | 0.91 (0.33) | 0.96 (0.24) | 0.81 (0.09)
  Month 60 (n=13,13,10) | 0.94 (0.29) | 0.97 (0.26) | 0.87 (0.10)
  Month 66 (n=12,14,10) | 1.05 (0.42) | 0.95 (0.26) | 0.84 (0.17)
  Month 72 (n=9,13,8) | 0.94 (0.24) | 0.95 (0.20) | 0.79 (0.12)
  Month 78 (n=0,13,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.95 (0.21) | 0.87 (0.10)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.94 (0.20) | 0.88 (0.12)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.91 (0.23) | 0.88 (0.14)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.90 (0.20) | 0.92 (0.12)
  Follow-Up (n=6,12,8) | 0.61 (0.27) | 0.91 (0.23) | 0.80 (0.28)

12. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With NODM, Definition 2 (NODM-2) by Visit
Description: Kaplan-Meier analysis of percentage of participants with NODM-2 by time to NODM-2 within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. NODM-2 was defined as an event experienced by a transplanted subject who meets any of the following criteria: (a) NODM-1; or (b) Symptoms of diabetes plus 2 casual serum glucose levels â‰¥200 mg/dL separated by at least approximately 24 hours. Casual was defined as any time of day without regard to time since last meal; or (c) Fasting serum glucose â‰¥126 mg/dL on 2 different occasions separated by at least approximately 24 hours. Fasting was defined as no caloric intake for at least 8 hours; or (d) 2-hour serum glucose â‰¥200 mg/dL during an OGTT (Oral Glucose Tolerance Test).
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants remaining at risk for the specified parameter at a given visit. Participants who had a history of diabetes at transplant were not included in the Kaplan-Meier analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 17 | 8 | 9
percentage of participants
  Day 1 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 1 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 3 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 6 (n=17,8,9) | 0.00 | 0.00 | 0.00
  Month 9 (n=16,7,9) | 5.88 | 12.50 | 0.00
  Month 12 (n=16,7,9) | 5.88 | 12.50 | 0.00
  Month 15 (n=16,7,9) | 5.88 | 12.50 | 0.00
  Month 18 (n=15,7,9) | 5.88 | 12.50 | 0.00
  Month 24 (n=15,7,9) | 5.88 | 12.50 | 0.00
  Month 30 (n=13,7,7) | 5.88 | 12.50 | 12.50
  Month 36 (n=13,7,7) | 5.88 | 12.50 | 12.50
  Month 42 (n=13,7,7) | 5.88 | 12.50 | 12.50
  Month 48 (n=12,7,7) | 5.88 | 12.50 | 12.50
  Month 54 (n=12,7,7) | 5.88 | 12.50 | 12.50
  Month 60 (n=11,7,7) | 5.88 | 12.50 | 12.50
  Month 66 (n=11,7,6) | 5.88 | 12.50 | 12.50
  Month 72 (n=6,7,6) | 14.44 | 12.50 | 12.50
  Month 78 (n=0,7,5) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 12.50 | 12.50
  Month 84 (n=0,7,5) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 12.50 | 12.50
  Month 90 (n=0,7,5) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 12.50 | 12.50
  Month 96 (n=0,7,5) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 12.50 | 12.50

13. Secondary Outcome: Total Cholesterol Levels by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mg/dL
  Month 9 (n=18,14,12) | 187.94 (44.81) | 233.71 (71.97) | 198.58 (40.95)
  Month 12 (n=16,14,12) | 180.31 (46.99) | 228.57 (64.34) | 210.08 (44.32)
  Month 15 (n=16,14,12) | 171.06 (40.13) | 208.79 (50.90) | 198.58 (30.80)
  Month 18 (n=18,14,12) | 173.28 (41.76) | 185.21 (45.99) | 192.00 (42.14)
  Month 24 (n=17,14,12) | 185.53 (62.85) | 188.64 (40.29) | 201.58 (47.21)
  Month 30 (n=14,14,10) | 175.43 (44.91) | 185.71 (37.82) | 198.30 (36.42)
  Month 36 (n=15,14,9) | 175.80 (42.49) | 174.86 (34.82) | 202.22 (31.25)
  Month 42 (n=15,14,9) | 179.87 (40.82) | 206.29 (78.76) | 187.67 (22.57)
  Month 48 (n=15,14,10) | 188.87 (64.11) | 195.79 (45.97) | 180.10 (38.08)
  Month 54 (n=14,14,10) | 184.86 (43.06) | 201.79 (51.39) | 183.70 (42.50)
  Month 60 (n=13,13,10) | 178.77 (50.20) | 184.23 (34.67) | 189.10 (56.48)
  Month 66 (n=12,14,10) | 188.25 (46.65) | 185.64 (46.46) | 172.20 (36.33)
  Month 72 (n=9,12,8) | 177.22 (43.21) | 186.42 (44.88) | 200.25 (57.28)
  Month 78 (n=0,13,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 191.85 (41.96) | 195.00 (48.57)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 192.42 (42.02) | 204.00 (36.43)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 185.92 (51.46) | 189.86 (30.62)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 183.27 (38.74) | 188.00 (18.89)
  Follow-Up (n=6,12,8) | 191.83 (41.84) | 185.58 (56.08) | 213.13 (40.70)

14. Secondary Outcome: Low-Density Lipoprotein (LDL) Levels by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mg/dL
  Month 9 (n=18,12,11) | 107.11 (37.14) | 138.83 (65.33) | 109.82 (32.60)
  Month 12 (n=16,14,12) | 102.75 (32.98) | 130.21 (50.51) | 119.42 (39.38)
  Month 15 (n=16,14,11) | 95.13 (28.34) | 117.29 (39.80) | 106.64 (26.98)
  Month 18 (n=18,14,12) | 95.94 (34.55) | 95.14 (37.28) | 104.42 (39.30)
  Month 24 (n=17,14,12) | 101.82 (48.27) | 99.29 (26.75) | 114.00 (38.82)
  Month 30 (n=14,14,10) | 97.93 (37.96) | 96.86 (26.09) | 115.50 (33.45)
  Month 36 (n=15,14,9) | 94.20 (34.49) | 90.29 (26.07) | 112.00 (27.83)
  Month 42 (n=15,13,9) | 100.27 (34.56) | 99.69 (36.08) | 102.11 (24.94)
  Month 48 (n=15,14,10) | 110.13 (55.46) | 107.07 (29.03) | 99.70 (34.56)
  Month 54 (n=14,13,10) | 108.36 (40.27) | 109.08 (32.78) | 96.50 (41.04)
  Month 60 (n=13,13,10) | 105.62 (42.86) | 101.00 (24.15) | 98.60 (44.67)
  Month 66 (n=12,13,10) | 109.83 (44.59) | 100.92 (33.67) | 91.90 (33.14)
  Month 72 (n=9,12,8) | 102.89 (43.96) | 100.00 (28.63) | 114.25 (46.57)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 103.25 (31.13) | 111.13 (41.46)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 103.92 (37.55) | 117.88 (32.73)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 101.92 (41.67) | 99.00 (23.93)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 93.82 (28.22) | 99.83 (30.30)
  Follow-Up (n=6,12,8) | 110.00 (49.37) | 102.42 (46.08) | 129.38 (39.71)

15. Secondary Outcome: High-Density Lipoprotein (HDL) Levels by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mg/dL
  Month 9 (n=18,14,12) | 54.83 (14.92) | 59.93 (14.38) | 52.58 (16.32)
  Month 12 (n=16,14,12) | 51.81 (18.82) | 62.07 (17.68) | 56.00 (16.99)
  Month 15 (n=16,14,12) | 51.31 (16.08) | 59.79 (16.37) | 53.08 (16.72)
  Month 18 (n=18,14,12) | 52.67 (17.07) | 59.29 (17.03) | 52.92 (15.17)
  Month 24 (n=17,14,12) | 53.76 (18.60) | 60.07 (17.09) | 55.17 (17.78)
  Month 30 (n=14,14,10) | 51.21 (16.83) | 59.29 (15.03) | 50.40 (9.29)
  Month 36 (n=15,14,9) | 53.13 (16.92) | 55.14 (15.42) | 56.44 (13.51)
  Month 42 (n=15,14,9) | 52.27 (14.40) | 56.57 (12.69) | 57.33 (12.23)
  Month 48 (n=15,14,10) | 49.67 (16.56) | 57.71 (17.73) | 50.10 (10.63)
  Month 54 (n=14,14,10) | 46.64 (13.28) | 60.07 (16.36) | 52.80 (12.27)
  Month 60 (n=13,13,10) | 45.23 (11.89) | 58.23 (15.69) | 58.30 (28.33)
  Month 66 (n=12,14,10) | 49.75 (15.72) | 56.57 (19.03) | 51.40 (13.92)
  Month 72 (n=9,12,8) | 46.67 (12.40) | 62.67 (15.25) | 48.38 (14.06)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 65.58 (18.75) | 49.38 (14.79)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 63.00 (17.79) | 46.38 (10.16)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 61.17 (14.94) | 49.57 (9.43)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 65.36 (18.78) | 52.00 (10.97)
  Follow-Up (n=6,12,8) | 55.67 (10.95) | 56.25 (15.78) | 45.38 (12.64)

16. Secondary Outcome: Ratio of Total Serum Cholesterol Level to HDL Level by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
ratio
  Month 9 (n=18,14,12) | 3.62 (1.05) | 4.09 (1.47) | 4.08 (1.34)
  Month 12 (n=16,14,12) | 3.72 (0.94) | 3.92 (1.40) | 4.03 (1.34)
  Month 15 (n=16,14,12) | 3.48 (0.78) | 3.66 (1.04) | 4.08 (1.33)
  Month 18 (n=18,14,12) | 3.50 (1.01) | 3.32 (1.03) | 3.88 (1.29)
  Month 24 (n=17,14,12) | 3.69 (1.28) | 3.35 (1.06) | 3.97 (1.43)
  Month 30 (n=14,14,10) | 3.70 (1.30) | 3.30 (0.99) | 4.03 (0.89)
  Month 36 (n=15,14,9) | 3.54 (1.23) | 3.35 (0.89) | 3.68 (0.61)
  Month 42 (n=15,14,9) | 3.63 (1.00) | 3.85 (1.82) | 3.35 (0.50)
  Month 48 (n=15,14,10) | 3.95 (1.04) | 3.59 (1.09) | 3.76 (1.20)
  Month 54 (n=14,14,10) | 4.17 (1.22) | 3.52 (1.14) | 3.64 (1.23)
  Month 60 (n=13,13,10) | 4.12 (1.18) | 3.32 (0.87) | 3.59 (1.20)
  Month 66 (n=12,14,10) | 3.99 (1.00) | 3.51 (1.08) | 3.50 (0.93)
  Month 72 (n=9,12,8) | 3.97 (1.08) | 3.05 (0.62) | 4.30 (1.31)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 3.06 (0.96) | 4.06 (0.89)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 3.22 (0.99) | 4.50 (0.96)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 3.14 (0.89) | 3.91 (0.74)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 2.97 (0.92) | 3.72 (0.69)
  Follow-Up (n=6,12,8) | 3.57 (1.06) | 3.45 (1.07) | 4.95 (1.27)

17. Secondary Outcome: Percentage of Participants With Ratio of Total Serum Cholesterol to Serum HDL Cholesterol <5 by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
percentage of participants
  Month 9 (n=18,14,12) | 94.4 | 71.4 | 66.7
  Month 12 (n=16,14,12) | 87.5 | 85.7 | 75.0
  Month 15 (n=16,14,12) | 93.8 | 92.9 | 66.7
  Month 18 (n=18,14,12) | 88.9 | 92.9 | 75.0
  Month 24 (n=17,14,12) | 88.2 | 85.7 | 66.7
  Month 30 (n=14,14,10) | 78.6 | 92.9 | 70.0
  Month 36 (n=15,14,9) | 86.7 | 100.0 | 100.0
  Month 42 (n=15,14,9) | 86.7 | 78.6 | 100.0
  Month 48 (n=15,14,10) | 86.7 | 92.9 | 80.0
  Month 54 (n=14,14,10) | 78.6 | 85.7 | 90.0
  Month 60 (n=13,13,10) | 69.2 | 92.3 | 80.0
  Month 66 (n=12,14,10) | 83.3 | 92.9 | 90.0
  Month 72 (n=9,12,8) | 88.9 | 100.0 | 75.0
  Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 87.5
  Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 91.7 | 50.0
  Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 100.0
  Month 96 (n=0,11,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 100.0
  Follow-Up (n=6,12,8) | 100.0 | 91.7 | 50.0

18. Secondary Outcome: Ratio of Serum LDL Level to HDL Level by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
ratio
  Month 9 (n=18,12,11) | 2.09 (0.84) | 2.42 (1.25) | 2.17 (0.82)
  Month 12 (n=16,14,12) | 2.14 (0.71) | 2.24 (0.98) | 2.31 (0.99)
  Month 15 (n=16,14,11) | 1.97 (0.62) | 2.07 (0.81) | 2.11 (0.74)
  Month 18 (n=18,14,12) | 1.98 (0.86) | 1.74 (0.80) | 2.10 (0.93)
  Month 24 (n=17,14,12) | 2.04 (0.94) | 1.78 (0.69) | 2.25 (0.98)
  Month 30 (n=14,14,10) | 2.09 (0.99) | 1.76 (0.69) | 2.36 (0.78)
  Month 36 (n=15,14,9) | 1.93 (0.92) | 1.75 (0.64) | 2.03 (0.49)
  Month 42 (n=15,13,9) | 2.06 (0.87) | 1.85 (0.81) | 1.82 (0.44)
  Month 48 (n=15,14,10) | 2.27 (0.85) | 1.99 (0.73) | 2.07 (0.80)
  Month 54 (n=14,13,10) | 2.48 (1.08) | 1.92 (0.81) | 1.92 (1.02)
  Month 60 (n=13,13,10) | 2.45 (0.99) | 1.86 (0.67) | 1.92 (0.98)
  Month 66 (n=12,13,10) | 2.34 (0.91) | 1.96 (0.85) | 1.88 (0.83)
  Month 72 (n=9,12,8) | 2.32 (1.00) | 1.66 (0.50) | 2.46 (1.04)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.72 (0.77) | 2.30 (0.80)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.80 (0.83) | 2.58 (0.69)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.74 (0.74) | 2.04 (0.50)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.56 (0.66) | 1.98 (0.69)
  Follow-up (n=6,12,8) | 2.09 (1.05) | 1.91 (0.82) | 3.03 (1.15)

19. Secondary Outcome: Percentage of Participants With Ratio of Serum LDL Cholesterol to Serum HDL Cholesterol <3.5 by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
percentage of participants
  Month 9 (n=18,12,11) | 94.4 | 75.0 | 90.9
  Month 12 (n=16,14,12) | 93.8 | 85.7 | 83.3
  Month 15 (n=16,14,11) | 100.0 | 92.9 | 100.0
  Month 18 (n=18,14,12) | 94.4 | 100.0 | 91.7
  Month 24 (n=17,14,12) | 94.1 | 100.0 | 91.7
  Month 30 (n=14,14,10) | 78.6 | 100.0 | 100.0
  Month 36 (n=15,14,9) | 93.3 | 100.0 | 100.0
  Month 42 (n=15,13,9) | 93.3 | 100.0 | 100.0
  Month 48 (n=15,14,10) | 93.3 | 92.9 | 90.0
  Month 54 (n=14,13,10) | 71.4 | 92.3 | 90.0
  Month 60 (n=13,13,10) | 76.9 | 100.0 | 90.0
  Month 66 (n=12,13,10) | 83.3 | 92.3 | 90.0
  Month 72 (n=9,12,8) | 88.9 | 100.0 | 75.0
  Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 87.5
  Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 87.5
  Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 100.0
  Month 96 (n=0,11,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.0 | 100.0
  Follow-Up (n=6,12,8) | 100.0 | 91.7 | 62.5

20. Secondary Outcome: Serum Triglyceride Levels by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mg/dL
  Month 9 (n=18,14,12) | 129.44 (53.45) | 205.07 (139.91) | 194.00 (128.60)
  Month 12 (n=16,14,12) | 129.19 (49.86) | 181.86 (107.49) | 173.00 (99.25)
  Month 15 (n=16,14,12) | 123.56 (52.90) | 158.93 (84.58) | 200.50 (122.75)
  Month 18 (n=18,14,12) | 123.44 (53.83) | 153.79 (79.29) | 173.08 (101.81)
  Month 24 (n=17,14,12) | 149.71 (86.56) | 146.50 (106.28) | 161.33 (83.95)
  Month 30 (n=14,14,10) | 131.07 (52.76) | 147.71 (84.28) | 162.30 (55.08)
  Month 36 (n=15,14,9) | 142.00 (68.44) | 147.14 (93.13) | 169.11 (79.39)
  Month 42 (n=15,14,9) | 136.60 (52.91) | 195.71 (156.42) | 141.22 (63.76)
  Month 48 (n=15,14,10) | 144.67 (70.99) | 155.07 (91.61) | 150.70 (106.82)
  Month 54 (n=14,14,10) | 150.14 (47.64) | 158.43 (115.94) | 170.90 (83.72)
  Month 60 (n=13,13,10) | 139.38 (71.94) | 125.23 (46.55) | 161.10 (93.01)
  Month 66 (n=12,14,10) | 143.42 (54.70) | 140.00 (117.56) | 145.30 (75.77)
  Month 72 (n=9,12,8) | 138.33 (59.14) | 118.33 (83.47) | 188.00 (72.59)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 104.42 (58.22) | 172.38 (53.73)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 127.17 (66.01) | 199.75 (84.79)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 113.75 (57.79) | 206.29 (83.17)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 119.64 (76.86) | 180.17 (93.92)
  Follow-Up (n=6,12,8) | 130.67 (63.87) | 134.50 (73.14) | 191.88 (83.21)

21. Secondary Outcome: Percentage of Participants Requiring Lipid-Lowering Agents by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 9 (n=18,14,13) | 38.9 | 64.3 | 53.8
  Month 12 (n=18,14,13) | 44.4 | 64.3 | 53.8
  Month 15 (n=18,14,12) | 44.4 | 71.4 | 50.0
  Month 18 (n=18,14,12) | 44.4 | 71.4 | 41.7
  Month 24 (n=17,14,12) | 47.1 | 71.4 | 58.3
  Month 30 (n=15,14,11) | 46.7 | 71.4 | 63.6
  Month 36 (n=15,14,11) | 46.7 | 71.4 | 72.7
  Month 42 (n=15,14,10) | 46.7 | 64.3 | 90.0
  Month 48 (n=15,14,10) | 46.7 | 64.3 | 90.0
  Month 54 (n=14,14,10) | 42.9 | 64.3 | 70.0
  Month 60 (n=13,14,10) | 38.5 | 64.3 | 80.0
  Month 66 (n=13,14,10) | 46.2 | 64.3 | 80.0
  Month 72 (n=9,14,9) | 44.4 | 64.3 | 88.9
  Month 78 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 61.5 | 87.5
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 61.5 | 87.5
  Month 90 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 58.3 | 87.5
  Month 96 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 58.3 | 100.0

22. Secondary Outcome: Percentage of Participants Requiring Anti-Hypertensive Medication by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 9 (n=18,14,13) | 83.3 | 85.7 | 92.3
  Month 12 (n=18,14,13) | 83.3 | 85.7 | 92.3
  Month 15 (n=18,14,12) | 83.3 | 85.7 | 91.7
  Month 18 (n=18,14,12) | 83.3 | 78.6 | 91.7
  Month 24 (n=17,14,12) | 82.4 | 85.7 | 91.7
  Month 30 (n=15,14,11) | 73.3 | 71.4 | 81.8
  Month 36 (n=15,14,10) | 73.3 | 71.4 | 90.0
  Month 42 (n=15,14,10) | 73.3 | 71.4 | 90.0
  Month 48 (n=15,14,10) | 73.3 | 71.4 | 90.0
  Month 54 (n=14,14,10) | 71.4 | 71.4 | 90.0
  Month 60 (n=13,14,10) | 69.2 | 71.4 | 90.0
  Month 66 (n=13,14,10) | 76.9 | 71.4 | 90.0
  Month 72 (n=9,14,9) | 77.8 | 71.4 | 88.9
  Month 78 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 69.2 | 87.5
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 69.2 | 75.0
  Month 90 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 66.7 | 75.0
  Month 96 (n=0,11,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 72.7 | 71.4

23. Secondary Outcome: Percentage of Participants Requiring Diabetes Agents (Oral Hypoglycemic Agents, Anti-Diabetic Agents, or Insulin) by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 9 (n=18,14,13) | 5.6 | 35.7 | 30.8
  Month 12 (n=18,14,12) | 5.6 | 35.7 | 33.3
  Month 15 (n=18,14,12) | 5.6 | 42.9 | 33.3
  Month 18 (n=18,14,12) | 11.1 | 42.9 | 33.3
  Month 24 (n=17,14,12) | 11.8 | 42.9 | 33.3
  Month 30 (n=15,14,11) | 13.3 | 42.9 | 27.3
  Month 36 (n=15,14,10) | 13.3 | 42.9 | 30.0
  Month 42 (n=15,14,10) | 13.3 | 42.9 | 30.0
  Month 48 (n=15,14,10) | 13.3 | 42.9 | 30.0
  Month 54 (n=14,14,10) | 14.3 | 42.9 | 30.0
  Month 60 (n=13,14,10) | 15.4 | 42.9 | 30.0
  Month 66 (n=13,14,10) | 15.4 | 42.9 | 30.0
  Month 72 (n=9,14,8) | 11.1 | 42.9 | 25.0
  Month 78 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 38.5 | 25.0
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 38.5 | 25.0
  Month 90 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 33.3 | 25.0
  Month 96 (n=0,11,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 36.4 | 16.7

24. Secondary Outcome: Epstein Barr Virus (EBV) Deooxyribonucleic Acid (DNA) Levels Determined Using Polymerase Chain Reaction (PCR) by Visit
Description: Calculated as number of copies per 500 mg DNA.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: number of copies/500 mg DNA
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 17 | 14 | 12
number of copies/500 mg DNA
  Month 9 (n=17,14,12) | 0.41 (1.46) | 1.00 (2.18) | 3.17 (3.30)
  Month 12 (n=17,14,12) | 0.12 (0.49) | 4.07 (11.89) | 8.42 (18.46)
  Month 15 (n=17,14,12) | 5.47 (22.05) | 6.71 (20.36) | 18.42 (24.27)
  Month 18 (n=17,13,12) | 0.59 (2.18) | 21.92 (56.56) | 21.50 (32.52)
  Month 24 (n=15,13,12) | 0.00 (0.00) | 10.38 (24.22) | 10.83 (25.90)
  Month 30 (n=13,14,10) | 2.15 (7.19) | 13.57 (31.74) | 23.80 (39.60)
  Month 36 (n=15,14,8) | 1.20 (3.19) | 8.64 (25.37) | 42.63 (110.49)
  Month 42 (n=14,12,9) | 0.57 (2.14) | 15.50 (19.10) | 17.00 (26.98)
  Month 48 (n=15,9,6) | 0.07 (0.26) | 17.00 (32.60) | 11.50 (21.42)
  Month 54 (n=14,14,10) | 0.64 (1.08) | 13.86 (26.40) | 6.30 (12.10)
  Month 60 (n=13,13,10) | 0.31 (0.63) | 11.46 (27.20) | 10.20 (20.86)
  Month 66 (n=10,13,9) | 0.40 (0.97) | 17.38 (26.83) | 31.11 (32.92)
  Month 72 (n=9,12,8) | 1.11 (3.33) | 11.08 (27.22) | 19.25 (41.80)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 10.08 (16.10) | 17.63 (42.28)
  Month 84 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 1.08 (1.51) | 10.88 (21.24)
  Month 90 (n=0,12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 2.92 (5.18) | 9.29 (20.69)
  Month 96 (n=0,9,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 5.67 (6.69) | 17.67 (23.11)

25. Secondary Outcome: Percentage of Participants With EBV DNA Determined Using PCR by Specific Cutoff Categories (in Number of Copies/PCR) and Visit
Description: EBV DNA PCR categories included 0, 1-50, 51-100, 101-1000, and >1000 copies/PCR.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96 and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 17 | 14 | 12
percentage of participants
  0: Month 9 (n=17,14,12) | 88.2 | 71.4 | 33.3
  0: Month 12 (n=17,14,12) | 94.1 | 64.3 | 33.3
  0: Month 15 (n=17,14,12) | 88.2 | 57.1 | 41.7
  0: Month 18 (n=17,13,12) | 88.2 | 53.8 | 41.7
  0: Month 24 (n=15,13,12) | 100.0 | 61.5 | 33.3
  0: Month 30 (n=13,14,10) | 84.6 | 42.9 | 30.0
  0: Month 36 (n=15,14,8) | 86.7 | 57.1 | 25.0
  0: Month 42 (n=14,12,9) | 92.9 | 33.3 | 22.2
  0: Month 48 (n=15,9,6) | 93.3 | 66.7 | 0
  0: Month 54 (n=14,14,10) | 57.1 | 50.0 | 30.0
  0: Month 60 (n=13,13,10) | 76.9 | 61.5 | 10.0
  0: Month 66 (n=10,13,9) | 80.0 | 38.5 | 0
  0: Month 72 (n=9,12,8) | 88.9 | 41.7 | 37.5
  0: Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 41.7 | 25.0
  0: Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 50.0 | 12.5
  0: Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 58.3 | 42.9
  0: Month 96 (n=0,9,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 33.3 | 33.3
  0: Follow-up (n=2,4,4) | 100.0 | 50.0 | 75.0
  1-50: Month 9 (n=17,14,12) | 11.8 | 28.6 | 66.7
  1-50: Month 12 (n=17,14,12) | 5.9 | 35.7 | 58.3
  1-50: Month 18 (n=17,13,12) | 11.8 | 30.8 | 41.7
  1-50: Month 24 (n=15,13,12) | 0 | 30.8 | 58.3
  1-50: Month 30 (n=13,14,10) | 15.4 | 50.0 | 60.0
  1-50: Month 36 (n=15,14,8) | 13.3 | 35.7 | 62.5
  1-50: Month 42 (n=14,12,9) | 7.1 | 58.3 | 66.7
  1-50: Month 48 (n=15,9,6) | 6.7 | 11.1 | 83.3
  1-50: Month 54 (n=14,14,10) | 42.9 | 42.9 | 70.0
  1-50: Month 60 (n=13,13,10) | 23.1 | 30.8 | 80.0
  1-50: Month 66 (n=10,13,9) | 20.0 | 46.2 | 55.6
  1-50: Month 72 (n=9,12,8) | 11.1 | 50.0 | 50.0
  1-50: Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 58.3 | 62.5
  1-50: Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 50.0 | 75.0
  1-50: Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 41.7 | 42.9
  1-50: Month 96 (n=0,9,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 66.7 | 50.0
  1-50: Follow-up (n=2,4,4) | 0 | 50.0 | 25.0
  51-100: Month 9 (n=17,14,12) | 0 | 0 | 0
  51-100: Month 12 (n=17,14,12) | 0 | 0 | 8.3
  51-100: Month 15 (n=17,14,12) | 5.9 | 7.1 | 8.3
  51-100: Month 18 (n=17,13,12) | 0 | 7.7 | 16.7
  51-100: Month 24 (n=15,13,12) | 0 | 7.7 | 8.3
  51-100: Month 30 (n=13,14,10) | 0 | 0 | 0
  51-100: Month 36 (n=15,14,8) | 0 | 7.1 | 0
  51-100: Month 42 (n=14,12,9) | 0 | 8.3 | 11.1
  51-100: Month 48 (n=15,9,6) | 0 | 22.2 | 16.7
  51-100: Month 54 (n=14,14,10) | 0 | 7.1 | 0
  51-100: Month 60 (n=13,13,10) | 0 | 7.7 | 10.0
  51-100: Month 66 (n=10,13,9) | 0 | 15.4 | 44.4
  51-100: Month 72 (n=9,12,8) | 0 | 8.3 | 0
  51-100: Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  51-100: Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 12.5
  51-100: Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 14.3
  51-100: Month 96 (n=0,9,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 16.7
  51-100: Follow-up (n=2,4,4) | 0 | 0 | 0
  101-1000: Month 9 (n=17,14,12) | 0 | 0 | 0
  101-1000: Month 12 (n=17,14,12) | 0 | 0 | 0
  101-1000: Month 15 (n=17,14,12) | 0 | 0 | 0
  101-1000: Month 18 (n=17,13,12) | 0 | 7.7 | 0
  101-1000: Month 24 (n=15,13,12) | 0 | 0 | 0
  101-1000: Month 30 (n=13,14,10) | 0 | 7.1 | 10.0
  101-1000: Month 36 (n=15,14,8) | 0 | 0 | 12.5
  101-1000: Month 42 (n=14,12,9) | 0 | 0 | 0
  101-1000: Month 48 (n=15,9,6) | 0 | 0 | 0
  101-1000: Month 54 (n=14,14,10) | 0 | 0 | 0
  101-1000: Month 60 (n=13,13,10) | 0 | 0 | 0
  101-1000: Month 66 (n=10,13,9) | 0 | 0 | 0
  101-1000: Month 72 (n=9,12,8) | 0 | 0 | 12.5
  101-1000: Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 12.5
  101-1000: Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  101-1000: Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  101-1000: Month 96 (n=0,9,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  101-1000: Follow-up (n=2,4,4) | 0 | 0 | 0
  >1000: Month 9 (n=17,14,12) | 0 | 0 | 0
  >1000: Month 12 (n=17,14,12) | 0 | 0 | 0
  >1000: Month 15 (n=17,14,12) | 0 | 0 | 0
  >1000: Month 18 (n=17,13,12) | 0 | 0 | 0
  >1000: Month 24 (n=15,13,12) | 0 | 0 | 0
  >1000: Month 30 (n=13,14,10) | 0 | 0 | 0
  >1000: Month 36 (n=15,14,8) | 0 | 0 | 0
  >1000: Month 42 (n=14,12,9) | 0 | 0 | 0
  >1000: Month 48 (n=15,9,6) | 0 | 0 | 0
  >1000: Month 54 (n=14,14,10) | 0 | 0 | 0
  >1000: Month 60 (n=13,13,10) | 0 | 0 | 0
  >1000: Month 66 (n=10,13,9) | 0 | 0 | 0
  >1000: Month 72 (n=9,12,8) | 0 | 0 | 0
  >1000: Month 78 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  >1000: Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  >1000: Month 90 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  >1000: Month 96 (n=0,9,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  >1000: Follow-up (n=2,4,4) | 0 | 0 | 0

26. Secondary Outcome: BK Virus (BKV) DNA Levels Determined Using PCR by Visit
Description: Calculated as number of copies per PCR. Per protocol, BKV DNA PCR was performed on tofacitinib-treated participants only.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: number of copies/PCR
Arm/Group | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 14 | 12
number of copies/PCR
  Month 9 (n=14,12) | 1.29 (4.53) | 1.58 (2.84)
  Month 12 (n=13,10) | 2.23 (3.81) | 0.10 (0.32)
  Month 15 (n=13,12) | 2.85 (7.66) | 0.75 (0.97)
  Month 18 (n=7,8) | 0.14 (0.38) | 0.38 (0.74)
  Month 24 (n=2,1) | 0.00 (0.00) | 0.00 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 30 (n=0,1) | NA (NA) — No participants were analyzed for the parameter at the specified timepoint. | 0.00 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 36 (n=5,4) | 15.80 (34.77) | 6.75 (13.50)
  Month 42 (n=11,7) | 0.64 (2.11) | 1.86 (4.49)
  Month 48 (n=9,6) | 8.33 (23.18) | 3.33 (8.16)
  Month 54 (n=13,10) | 4.54 (14.66) | 1.40 (3.78)
  Month 60 (n=13,7) | 15.85 (41.81) | 0.86 (2.27)
  Month 66 (n=13,8) | 6.15 (21.00) | 0.00 (0.00)
  Month 72 (n=10,7) | 1.00 (2.83) | 0.14 (0.38)
  Month 78 (n=9,7) | 0.56 (1.13) | 0.14 (0.38)
  Month 84 (n=10,7) | 0.60 (1.90) | 0.14 (0.38)
  Month 90 (n=9,4) | 0.56 (1.67) | 0.00 (0.00)
  Month 96 (n=9,3) | 1.11 (2.67) | 0.00 (0.00)
  Follow-up (n=3,2) | 0.00 (0.00) | 0.50 (0.71)

27. Secondary Outcome: Percentage of Participants With BKV DNA Determined Using PCR by Specific Cutoff Categories (in Number of Copies/PCR) and Visit
Description: Cutoff categories for BKV DNA were 0-199 and ≥200 copies/PCR. Per protocol, BKV DNA PCR was performed on tofacitinib-treated participants only.
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 14 | 12
percentage of participants
  0-199: Month 9 (n=14,12) | 100.0 | 100.0
  0-199: Month 12 (n=13,10) | 100.0 | 100.0
  0-199: Month 15 (n=13,12) | 100.0 | 100.0
  0-199: Month 18 (n=7,8) | 100.0 | 100.0
  0-199: Month 24 (n=2,1) | 100.0 | 100.0
  0-199: Month 30 (n=0,1) | 0 | 100.0
  0-199: Month 36 (n=5,4) | 100.0 | 100.0
  0-199: Month 42 (n=11,7) | 100.0 | 100.0
  0-199: Month 48 (n=9,6) | 100.0 | 100.0
  0-199: Month 54 (n=13,10) | 100.0 | 100.0
  0-199: Month 60 (n=13,7) | 100.0 | 100.0
  0-199: Month 66 (n=13,8) | 100.0 | 100.0
  0-199: Month 72 (n=10,7) | 100.0 | 100.0
  0-199: Month 78 (n=9,7) | 100.0 | 100.0
  0-199: Month 84 (n=10,7) | 100.0 | 100.0
  0-199: Month 90 (n=9,4) | 100.0 | 100.0
  0-199: Month 96 (n=9,3) | 100.0 | 100.0
  0-199: Follow-up (n=3,2) | 100.0 | 100.0
  ≥200: Month 9 (n=14,12) | 0 | 0
  ≥200: Month 12 (n=13,10) | 0 | 0
  ≥200: Month 15 (n=13,12) | 0 | 0
  ≥200: Month 18 (n=7,8) | 0 | 0
  ≥200: Month 24 (n=2,1) | 0 | 0
  ≥200: Month 30 (n=0,1) | 0 | 0
  ≥200: Month 36 (n=5,4) | 0 | 0
  ≥200: Month 42 (n=11,7) | 0 | 0
  ≥200: Month 48 (n=9,6) | 0 | 0
  ≥200: Month 54 (n=13,10) | 0 | 0
  ≥200: Month 60 (n=13,7) | 0 | 0
  ≥200: Month 66 (n=13,8) | 0 | 0
  ≥200: Month 72 (n=10,7) | 0 | 0
  ≥200: Month 78 (n=9,7) | 0 | 0
  ≥200: Month 84 (n=10,7) | 0 | 0
  ≥200: Month 90 (n=9,4) | 0 | 0
  ≥200: Month 96 (n=9,3) | 0 | 0
  ≥200: Follow-up (n=3,2) | 0 | 0

28. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Cytomegalovirus (CMV) Disease by Visit
Description: Kaplan-Meier analysis of percentage of participants with CMV disease within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. CMV disease was an adverse event associated with the preferred term 'CMV infection'.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: Safety population; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 3 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 6 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 9 (n=18,13,12) | 0.00 | 7.14 | 7.69
  Month 12 (n=18,13,12) | 0.00 | 7.14 | 7.69
  Month 15 (n=17,13,12) | 5.56 | 7.14 | 7.69
  Month 18 (n=16,13,12) | 5.56 | 7.14 | 7.69
  Month 24 (n=16,13,12) | 5.56 | 7.14 | 7.69
  Month 30 (n=14,13,11) | 5.56 | 7.14 | 7.69
  Month 36 (n=14,13,11) | 5.56 | 7.14 | 7.69
  Month 42 (n=14,13,10) | 5.56 | 7.14 | 7.69
  Month 48 (n=13,13,10) | 5.56 | 7.14 | 7.69
  Month 54 (n=13,13,10) | 5.56 | 7.14 | 7.69
  Month 60 (n=12,13,10) | 5.56 | 7.14 | 7.69
  Month 66 (n=12,13,9) | 5.56 | 7.14 | 7.69
  Month 72 (n=5,13,8) | 5.56 | 7.14 | 7.69
  Month 78 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 7.69
  Month 84 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 7.69
  Month 90 (n=0,12,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 7.69
  Month 96 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 7.69

29. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With First Biopsy-Proven Chronic Allograft Nephropathy (BPCAN) by Visit
Description: Kaplan-Meier analysis of percentage of participants with first BPCAN by time to first BPCAN within 96 months post-transplant. BPCAN was defined as chronic allograft nephropathy (Category 5 of the Banff Classification), based on the assessment of the renal allograft biopsy by a central, blinded pathologist. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. Includes BPCAN diagnosed on biopsies done for cause and ready by the central pathologist.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: FAS; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 3 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 6 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 9 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 12 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 15 (n=18,14,12) | 0.00 | 0.00 | 7.69
  Month 18 (n=17,14,12) | 0.00 | 0.00 | 7.69
  Month 24 (n=17,14,11) | 0.00 | 0.00 | 15.38
  Month 30 (n=15,14,10) | 0.00 | 0.00 | 15.38
  Moth 36 (n=15,14,10) | 0.00 | 0.00 | 15.38
  Month 42 (n=15,14,9) | 0.00 | 0.00 | 15.38
  Month 48 (n=14,14,9) | 0.00 | 0.00 | 15.38
  Month 54 (n=14,14,9) | 0.00 | 0.00 | 15.38
  Month 60 (n=13,14,9) | 0.00 | 0.00 | 15.38
  Month 66 (n=13,14,8) | 0.00 | 0.00 | 15.38
  Month 72 (n=6,14,7) | 0.00 | 0.00 | 15.38
  Month 78 (n=0,14,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38
  Month 84 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38
  Month 90 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38
  Month 96 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 15.38

30. Secondary Outcome: Cumulative Percentage of Participants With a First Antibody-Mediated Rejection or First BPAR
Description: Antibody-mediated rejection is defined as Category 2 and BPAR is defined as Category 4 of the Banff Classification, based on the assessment of the renal allograft biopsy by a central, blinded pathologist. Acute humoral rejection was categorized as Grades I, II, III and acute/active cellular rejection was categorized as Grades IA, IB, IIA, IIB, and III. Only participants with first BPAR were included.
Time Frame: Months 12, 18, 24, 36, 48, 60, 72, 84, 96, and Follow-Up (Month 98)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 12 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 18 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 24 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 36 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 48 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 60 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 72 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 84 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 96 Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Follow-up Antibody-mediated rejection (n=18,14,13) | 0 | 0 | 0
  Month 12 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 18 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 24 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 36 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 48 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 60 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 72 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 84 BPAR (n=18,14,13) | 0 | 0 | 0
  Month 96 BPAR (n=18,14,13) | 0 | 0 | 0
  Follow-up BPAR (n=18,14,13) | 0 | 0 | 0

31. Secondary Outcome: Cumulative Percentage of Participants With Ordered Categorical Severity of First BPCAN
Description: Ordered categorical severity of first BPCAN was classified according to the Banff Classification. Grade I: mild, grade II: moderate and grade III: severe interstitial fibrosis and tubular atrophy/loss. (Racusen et al: The Banff classification, 1999).
Time Frame: Months 12, 18, 24, 36, 48, 60, 72, 84, and 96
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Month 12: Grade I | 0 | 0 | 0
  Month 12: Grade II | 0 | 0 | 0
  Month 12: Grade III | 0 | 0 | 0
  Month 18: Grade I | 0 | 0 | 0
  Month 18: Grade II | 0 | 0 | 7.7
  Month 18: Grade III | 0 | 0 | 0
  Month 24: Grade I | 0 | 0 | 0
  Month 24: Grade II | 0 | 0 | 7.7
  Month 24: Grade III | 0 | 0 | 0
  Month 36: Grade I | 0 | 0 | 0
  Month 36: Grade II | 0 | 0 | 7.7
  Month 36: Grade III | 0 | 0 | 0
  Month 48: Grade I | 0 | 0 | 0
  Month 48: Grade II | 0 | 0 | 7.7
  Month 48: Grade III | 0 | 0 | 0
  Month 60: Grade I | 0 | 0 | 0
  Month 60: Grade II | 0 | 0 | 7.7
  Month 60: Grade III | 0 | 0 | 0
  Month 72: Grade I | 0 | 0 | 0
  Month 72: Grade II | 0 | 0 | 7.7
  Month 72: Grade III | 0 | 0 | 0
  Month 84: Grade I | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  Month 84: Grade II | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 7.7
  Month 84: Grade III | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  Month 96: Grade I | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0
  Month 96: Grade II | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 7.7
  Month 96: Grade III | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0 | 0

32. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Efficacy Failure by Visit
Description: Kaplan-Meier analysis of percentage of participants with efficacy failure by time to first efficacy failure within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. Efficacy failure was defined as first occurrence of BPAR, death, or graft loss.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: FAS; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=17,14,13) | 5.56 | 0.00 | 0.00
  Month 3 (n=17,14,11) | 5.56 | 0.00 | 15.38
  Month 6 (n=17,14,11) | 5.56 | 0.00 | 15.38
  Month 9 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 12 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 15 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 18 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 24 (n=16,14,11) | 11.11 | 0.00 | 15.38
  Month 30 (n=14,14,10) | 11.11 | 0.00 | 15.38
  Month 36 (n=14,14,10) | 11.11 | 0.00 | 15.38
  Month 42 (n=14,14,9) | 11.11 | 0.00 | 15.38
  Month 48 (n=13,14,9) | 11.11 | 0.00 | 15.38
  Month 54 (n=13,14,9) | 11.11 | 0.00 | 15.38
  Month 60 (n=12,14,9) | 11.11 | 0.00 | 15.38
  Month 66 (n=12,14,8) | 11.11 | 0.00 | 15.38
  Month 72 (n=5,14,7) | 11.11 | 0.00 | 25.96
  Month 78 (n=0,14,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 0.00 | 25.96
  Month 84 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 25.96
  Month 90 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 25.96
  Month 96 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 25.96

33. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Graft Survival by Visit
Description: Kaplan-Meier analysis of percentage of participants with graft survival by time to graft loss within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. Graft loss was defined as graft nephrectomy, retransplantation, return to dialysis for â‰¥6 consecutive weeks, or death.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: FAS; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 1 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 3 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 6 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 9 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 12 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 15 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 18 (n=17,14,13) | 100.00 | 100.00 | 100.00
  Month 24 (n=17,14,13) | 100.00 | 100.00 | 100.00
  Month 30 (n=15,14,12) | 100.00 | 100.00 | 100.00
  Month 36 (n=15,14,12) | 100.00 | 100.00 | 100.00
  Month 42 (n=15,14,11) | 100.00 | 100.00 | 100.00
  Month 48 (n=14,14,11) | 100.00 | 100.00 | 100.00
  Month 54 (n=14,14,11) | 100.00 | 100.00 | 100.00
  Month 60 (n=13,14,11) | 100.00 | 100.00 | 100.00
  Month 66 (n=13,14,10) | 100.00 | 100.00 | 100.00
  Month 72 (n=6,14,9) | 100.00 | 100.00 | 90.00
  Month 78 (n=0,14,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.00 | 90.00
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 92.86 | 90.00
  Month 90 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 92.86 | 90.00
  Month 96 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 92.86 | 90.00

34. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants Surviving by Visit
Description: Kaplan-Meier analysis of percentage of participants surviving by time to event (death) within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: FAS; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 1 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 3 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 6 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 9 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 12 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 15 (n=18,14,13) | 100.00 | 100.00 | 100.00
  Month 18 (n=17,14,13) | 100.00 | 100.00 | 100.00
  Month 24 (n=17,14,13) | 100.00 | 100.00 | 100.00
  Month 30 (n=15,14,12) | 100.00 | 100.00 | 100.00
  Month 36 (n=15,14,12) | 100.00 | 100.00 | 100.00
  Month 42 (n=15,14,11) | 100.00 | 100.00 | 100.00
  Month 48 (n=14,14,11) | 100.00 | 100.00 | 100.00
  Month 54 (n=14,14,11) | 100.00 | 100.00 | 100.00
  Month 60 (n=13,14,11) | 100.00 | 100.00 | 100.00
  Month 66 (n=13,14,10) | 100.00 | 100.00 | 100.00
  Month 72 (n=6,14,9) | 100.00 | 100.00 | 90.00
  Month 78 (n=0,14,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 100.00 | 90.00
  Month 84 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 92.86 | 90.00
  Month 90 (n=0,13,8) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 92.86 | 90.00
  Month 96 (n=0,12,7) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 92.86 | 90.00

35. Secondary Outcome: Kaplan-Meier Analysis of Percentage of Participants With Rejection by Visit
Description: Kaplan-Meier analysis of percentage of participants with rejection by time to rejection within 96 months post-transplant. Time was defined from the date of first dose of study drug in Study A3921009 to the date of first occurrence of the event, censored at the day of the last visit or Day 2980 (the maximum scheduled day for follow-up 98 month), whichever comes earlier. Rejection was defined as first occurrence of BPAR, antibody-mediated rejection or suspicious for acute rejection. This included biopsies read by the central pathologist.
Time Frame: Day 1 and Months 1, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96
Population: FAS; n=number of participants remaining at risk for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 13
percentage of participants
  Day 1 (n=18,14,13) | 0.00 | 0.00 | 0.00
  Month 1 (n=17,13,13) | 5.56 | 7.14 | 0.00
  Month 3 (n=17,13,11) | 5.56 | 7.14 | 15.38
  Month 6 (n=17,13,11) | 5.56 | 7.14 | 15.38
  Month 9 (n=16,13,11) | 11.11 | 7.14 | 15.38
  Month 12 (n=16,13,11) | 11.11 | 7.14 | 15.38
  Month 15 (n=16,13,11) | 11.11 | 7.14 | 15.38
  Month 18 (n=16,13,11) | 11.11 | 7.14 | 15.38
  Month 24 (n=16,13,11) | 11.11 | 7.14 | 15.38
  Month 30 (n=14,13,10) | 11.11 | 7.14 | 15.38
  Month 36 (n=14,13,10) | 11.11 | 7.14 | 15.38
  Month 42 (n=14,13,9) | 11.11 | 7.14 | 15.38
  Month 48 (n=13,13,9) | 11.11 | 7.14 | 15.38
  Month 54 (n=13,13,9) | 11.11 | 7.14 | 15.38
  Month 60 (n=12,13,9) | 11.11 | 7.14 | 15.38
  Month 66 (n=12,13,8) | 11.11 | 7.14 | 15.38
  Month 72 (n=5,13,6) | 11.11 | 7.14 | 27.47
  Month 78 (n=0,13,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 27.47
  Month 84 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 27.47
  Month 90 (n=0,12,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 27.47
  Month 96 (n=0,11,6) | NA — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.14 | 27.47

36. Secondary Outcome: Absolute Cluster of Differentiation (CD) 8+, CD19+, CD4+, and CD56+ Flouresence Activated Cell Sorting (FACS) Counts (Cells/uL) by Visit
Time Frame: Months 12 and 24
Population: Safety population
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 15 | 14 | 12
cells/uL
  CD8+: Month 12 | 284.67 (218.43) | 207.43 (97.19) | 232.33 (110.61)
  CD8+: Month 24 | 318.20 (183.85) | 224.36 (194.45) | 238.08 (172.46)
  CD19+: Month 12 | 197.53 (209.42) | 169.64 (97.97) | 127.42 (67.08)
  CD19+: Month 24 | 144.47 (116.77) | 125.86 (79.56) | 85.08 (51.02)
  CD4+: Month 12 | 612.80 (339.75) | 634.86 (280.75) | 565.00 (222.61)
  CD4+: Month 24 | 599.13 (216.61) | 462.00 (295.73) | 457.83 (202.29)
  CD56+: Month 12 | 152.67 (198.33) | 50.14 (43.96) | 35.58 (30.60)
  CD56+: Month 24 | 135.27 (145.25) | 77.86 (107.37) | 59.17 (69.31)

37. Secondary Outcome: Hemoglobin A1c (HbA1c) Levels by Visit
Time Frame: Months 12, 24, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96 and Follow-up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: % HbA1c
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 16 | 14 | 12
% HbA1c
  Month 12 (n=16,14,12) | 5.65 (0.69) | 6.84 (2.04) | 6.02 (0.82)
  Month 24 (n=16,14,12) | 5.63 (0.68) | 7.12 (2.20) | 6.28 (1.24)
  Month 36 (n=15,14,8) | 5.75 (1.21) | 7.19 (2.44) | 6.56 (1.35)
  Month 42 (n=15,14,9) | 5.81 (1.08) | 7.40 (2.56) | 6.68 (1.64)
  Month 48 (n=15,14,10) | 6.03 (1.23) | 7.25 (2.37) | 6.25 (0.82)
  Month 54 (n=14,14,10) | 6.39 (1.86) | 7.25 (1.94) | 6.43 (1.28)
  Month 60 (n=12,12,10) | 6.18 (1.11) | 7.03 (1.75) | 6.48 (1.47)
  Month 66 (n=12,14,10) | 6.13 (1.29) | 6.99 (1.82) | 6.52 (1.59)
  Month 72 (n=9,12,8) | 6.31 (1.72) | 6.93 (1.88) | 6.29 (1.38)
  Month 78 (n=12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 7.27 (2.52) | 6.43 (1.98)
  Month 84 (n=12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 6.66 (1.85) | 5.99 (1.00)
  Month 90 (n=12,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 6.38 (1.80) | 6.54 (2.08)
  Month 96 (n=11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 6.32 (1.42) | 6.77 (2.44)
  Follow-up (n=3,13,6) | 6.50 (2.00) | 6.65 (1.76) | 7.22 (2.71)

38. Secondary Outcome: Homeostatic Model Assessment (HOMA)-%B by Visit
Description: HOMA-%B = (20 times [*] fasting serum insulin) divided by (/) (fasting serum glucose minus [-] 3.5). HOMA-%B was only performed in participants who were non-diabetic prior to kidney transplantation and who did not require treatment with oral hypoglycemic agents, anti-diabetic agents, and/or insulin prior to the time of measurements.
Time Frame: Months 12 and 24
Population: Safety population; n=number of participants who were eligible for OGTT and had data (non-missing) at that particular visit.
Measure: Mean (Standard Deviation); unit: %B
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 9 | 6 | 5
%B
  Month 12 (n=8,6,5) | 204.67 (195.58) | 142.23 (95.06) | 194.65 (131.16)
  Month 24 (n=9,6,5) | 224.75 (333.49) | 138.10 (89.84) | 165.38 (68.73)

39. Secondary Outcome: Ratio of Fasting Serum Proinsulin (Pmol/L) to Insulin (Pmol/L) by Visit
Description: Measured only in participants who were non-diabetic prior to kidney transplantation and who did not require treatment with oral hypoglycemic agents, anti-diabetic agents, and/or insulin prior to the time of measurement.
Time Frame: Months 12 and 24
Population: Safety population; n=number of participants eligible for OGTT and had data (non-missing) at that particular visit.
Measure: Mean (Standard Deviation); unit: ratio of serum proinsulin to insulin
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 5 | 4 | 2
ratio of serum proinsulin to insulin
  Month 12 (n=5,3,3) | 0.15 (0.07) | 0.32 (0.04) | 0.40 (0.31)
  Month 24 (n=3,4,2) | 0.64 (0.42) | 0.30 (0.20) | 0.22 (0.04)

40. Secondary Outcome: Area Under the Curve (AUC) of Serum Glucose (mg*h/dL) Measured During Oral Glucose Tolerance Test (OGTT) by Visit
Description: Only performed in participants who were non-diabetic prior to kidney transplantation and who did not require treatment with oral hypoglycemic agents, anti-diabetic agents, and/or insulin.
Time Frame: Months 12 and 24
Population: Safety population; n=number of participants eligible for OGTT with data (non-missing) at that particular visit.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 12 | 8 | 6
mg*h/dL
  Month 12 (n=10,6,6) | 234.78 (58.78) | 254.25 (72.34) | 281.54 (52.39)
  Month 24 (n=12,8,5) | 230.10 (56.41) | 236.94 (92.98) | 281.90 (100.76)

41. Secondary Outcome: AUC of Serum Insulin (microU*h/mL) Measured During OGTT by Visit
Description: The OGTT was performed only in participants who were non-diabetic prior to kidney transplantation and who did not require treatment with oral hypoglycemic agents, anti-diabetic agents, and/or insulin.
Time Frame: Months 12 and 24
Population: Safety population: n=number of participants who were eligible for OGTT and had data (non-mising) at that particular visit.
Measure: Mean (Standard Deviation); unit: microU*h/mL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 10 | 6 | 6
microU*h/mL
  Month 12 (n=10,6,6) | 85.05 (37.57) | 99.96 (54.22) | 153.46 (92.11)
  Month 24 (n=8,6,5) | 79.84 (42.65) | 130.63 (48.07) | 181.70 (155.32)

42. Secondary Outcome: HOMA Insulin Resistance (IR) by Visit
Description: HOMA-IR=fasting serum insulin*fasting serum glucose/22.5. Measurement only performed in participants who were non-diabetic prior to kidney transplantation and who do not require treatment with oral hypoglycemic agents, anti diabetic agents, and/or insulin prior to the time of measurement.
Time Frame: Months 12 and 24
Population: Safety population; n=number of participants who were eligible for OGTT and had data (non-mising) at that particular visit.
Measure: Mean (Standard Deviation); unit: HOMA-IR
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 9 | 6 | 5
HOMA-IR
  Month 12 (n=8,6,5) | 2.55 (1.49) | 2.24 (1.85) | 2.54 (1.51)
  Month 24 (n=9,6,5) | 2.67 (2.76) | 9.01 (18.37) | 2.68 (1.19)

43. Secondary Outcome: Fasting Serum Glucose Levels (mg/dL) by Visit
Time Frame: Months 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-Up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 18 | 14 | 12
mg/dL
  Month 9 (n=18,14,10) | 96.89 (18.78) | 115.14 (42.16) | 97.90 (19.44)
  Month 12 (n=17,14,12) | 103.00 (26.25) | 133.79 (51.07) | 102.75 (35.70)
  Month 15 (n=17,13,11) | 95.41 (20.99) | 128.08 (85.36) | 99.18 (33.34)
  Month 18 (n=18,14,12) | 94.72 (21.38) | 117.93 (51.81) | 112.50 (48.45)
  Month 24 (n=17,14,12) | 113.71 (32.54) | 115.64 (45.68) | 122.25 (33.94)
  Month 30 (n=14,14,10) | 102.50 (29.02) | 137.86 (77.07) | 140.00 (79.88)
  Month 36 (n=15,14,9) | 108.20 (39.01) | 128.00 (54.34) | 143.33 (76.69)
  Month 42 (n=15,14,9) | 104.47 (30.92) | 113.71 (47.34) | 109.56 (34.93)
  Month 48 (n=15,14,10) | 112.93 (49.35) | 123.29 (77.74) | 98.00 (13.80)
  Month 54 (n=12,14,10) | 126.58 (81.04) | 119.21 (50.14) | 116.30 (69.12)
  Month 60 (n=12,12,10) | 107.08 (22.95) | 136.17 (68.68) | 111.70 (34.86)
  Month 66 (n=10,13,10) | 111.90 (36.39) | 143.77 (103.15) | 112.90 (48.43)
  Month 72 (n=9,13,7) | 100.44 (39.41) | 117.69 (61.22) | 127.43 (74.82)
  Month 78 (n=0,12,8) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 131.67 (66.25) | 98.50 (30.07)
  Month 84 (n=0,12,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 139.50 (86.88) | 112.50 (50.12)
  Month 90 (n=0,11,7) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 114.55 (33.39) | 96.43 (16.83)
  Month 96 (n=0,11,6) | NA (NA) — The tacrolimus treatment group was discontinued after Month 72, thus no participants were analyzed for this parameter at this timepoint. | 154.64 (115.73) | 100.33 (15.65)
  Follow-up (n=6,10,7) | 112.17 (42.96) | 126.30 (75.84) | 98.86 (31.73)

44. Secondary Outcome: Tofacitinib Concentrations in Plasma (ng/mL) by Visit
Time Frame: Months 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, and Follow-up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 14 | 12
ng/mL
  Month 9, predose (n=13,11) | 40.97 (46.65) | 12.38 (7.60)
  Month 9, 0.5 hours postdose (n=0,1) | NA (NA) — No participants were analyzed for the parameter at the specified timepoint. | 24.00 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 12, predose (n=13,12) | 14.75 (10.44) | 32.86 (46.50)
  Month 12, 1 hour postdose (n=1,0) | 51.50 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | NA (NA) — No participants were analyzed for the parameter at the specified timepoint.
  Month 18, predose (n=12,10) | 13.77 (10.60) | 7.84 (7.37)
  Month 18, 0.5 hours postdose (n=0,1) | NA (NA) — No participants were analyzed for the parameter at the specified timepoint. | 86.30 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 18, 1 hour postdose (n=0,1) | NA (NA) — No participants were analyzed for the parameter at the specified timepoint. | 80.70 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 24, predose (n=14,12) | 15.43 (11.14) | 28.15 (45.77)
  Month 24, 0.5 hours postdose (n=5,2) | 28.02 (4.44) | 96.30 (32.10)
  Month 24, 1 hour postdose (n=6,3) | 40.88 (9.28) | 72.33 (35.80)
  Month 30, predose (n=14,9) | 6.53 (5.37) | 16.18 (19.46)
  Month 30, 0.5 hours postdose (n=5,2) | 51.44 (26.39) | 54.95 (16.05)
  Month 30, 1 hour postdose (n=5,2) | 57.78 (10.90) | 98.45 (30.48)
  Month 36, predose (n=14,8) | 6.73 (4.49) | 13.28 (9.88)
  Month 42, predose (n=14, 8) | 19.70 (29.98) | 22.01 (13.71)
  Month 48, predose (n=12,9) | 9.71 (6.51) | 15.54 (7.33)
  Month 48, 0.5 hours postdose (n=1,1) | 1.00 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | 55.70 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 48, 1 hour postdose (n=1,0) | 56.60 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | NA (NA) — No participants were analyzed for the parameter at the specified timepoint.
  Month 54, predose (n=14,10) | 15.99 (14.97) | 24.74 (41.68)
  Month 60, predose (n=11,10) | 10.69 (9.62) | 15.03 (10.78)
  Month 60, 0.5 hours postdose (n=1,0) | 41.10 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | NA (NA) — No participants were analyzed for the parameter at the specified timepoint.
  Month 66, predose (n=11,10) | 14.64 (15.04) | 22.78 (18.11)
  Month 66, 0.5 hours postdose (n=1,2) | 27.70 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | 29.75 (18.17)
  Month 66, 1 hour postdose (n=1,1) | 18.90 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | 29.10 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 72, predose (n=9,7) | 10.07 (14.63) | 20.43 (20.53)
  Month 78, predose (n=10,8) | 4.13 (3.00) | 18.94 (18.48)
  Month 84, predose (n=11,5) | 21.46 (37.92) | 11.93 (6.59)
  Month 90, predose (n=10,5) | 6.91 (7.88) | 13.28 (9.78)
  Month 90, 0.5 hours postdose (n=0,1) | NA (NA) — No participants were analyzed for the parameter at the specified timepoint. | 17.70 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Month 96, predose (n=10,6) | 21.07 (39.16) | 31.97 (24.39)
  Follow-up, predose (n=1,1) | 16.00 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed. | 1.00 (NA) — No measure of dispersion could be determined as only 1 participant was analyzed.
  Follow-up, 0.5 hours postdose (n=2,4) | 2.57 (2.23) | 5.39 (5.28)

45. Secondary Outcome: Trough Levels of Tacrolimus (ng/mL) by Visit
Time Frame: Months 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, and 72 and Follow-up (Month 98)
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus
Number analyzed (Participants) | 16
ng/mL
  Month 9 (n=16) | 7.00 (1.55)
  Month 12 (n=10) | 9.50 (5.08)
  Month 18 (n=17) | 8.00 (2.81)
  Month 24 (n=9) | 8.78 (3.93)
  Month 30 (n=12) | 6.17 (2.55)
  Month 36 (n=15) | 6.87 (2.26)
  Month 42 (n=13) | 7.08 (1.85)
  Month 48 (n=15) | 8.07 (2.96)
  Month 54 (n=1) | 10.00 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint.
  Month 60 (n=12) | 6.58 (3.78)
  Month 72 (n=8) | 7.13 (1.64)
  Follow-up (n=1) | 8.00 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint.

46. Secondary Outcome: Short-Form 36 Version 2 (SF-36 v2) Mental Component Summary (MCS) and Physical Component Summary (PCS) Scores by Visit and Scale
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component scores (PCS and MCS). Total of 11 variables were analyzed (8 subscales, 2 composite subscales and Question 2 "how would you rate your health in general now?" (range 1= better, 5= worst). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety Population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 16 | 13 | 12
score on a scale
  PCS: Month 12 (n=12,13,9) | 54.33 (7.83) | 51.71 (10.22) | 46.05 (8.70)
  PCS: Month 18 (n=15,12,10) | 53.76 (8.18) | 50.67 (10.48) | 46.89 (9.61)
  PCS: Month 24 (n=16,13,12) | 50.82 (9.33) | 52.17 (8.06) | 48.85 (7.40)
  MCS: Month 12 (n=12,13,9) | 53.39 (7.93) | 50.83 (11.12) | 54.08 (10.32)
  MCS: Month 18 (n=15,12,10) | 49.70 (10.59) | 53.92 (10.61) | 51.44 (12.21)
  MCS: Month 24 (n=16,13,12) | 50.70 (9.40) | 55.61 (6.00) | 52.14 (8.89)

47. Secondary Outcome: Change From Baseline in SF-36 v2 MCS and PCS Scores by Visit and Scale
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as PCS and MCS. Total of 11 variables were analyzed (8 subscales, 2 composite subscales and Question 2 "how would you rate your health in general now?" (range 1= better, 5= worst). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Negative change from baseline represented improvement.
Time Frame: Baseline, Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 13 | 11 | 10
scores on a scale
  PCS: Month 12 (n=12,11,9) | 9.61 (6.21) | 6.23 (8.75) | 3.20 (10.71)
  PCS: Month 18 (n=13,9,8) | 10.82 (6.29) | 5.65 (7.84) | 2.76 (10.26)
  PCS: Month 24 (n=13,10,10) | 9.67 (5.55) | 7.09 (7.25) | 4.36 (8.60)
  MCS: Month 12 (n=12,11,9) | 6.86 (7.35) | 5.03 (13.29) | 13.70 (12.32)
  MCS: Month 18 (n=13,9,8) | 1.91 (14.71) | 9.54 (9.53) | 8.57 (13.96)
  MCS: Month 24 (n=13,10,10) | 2.99 (11.63) | 10.05 (12.55) | 9.59 (15.22)

48. Secondary Outcome: SF-36 v2 Subscale Scores by Visit
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as PCS and MCS. Total of 11 variables were analyzed (8 subscales, 2 composite subscales and Question 2 "how would you rate your health in general now?" (range 1= better, 5= worst). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety Population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 16 | 13 | 12
scores on a scale
  Phys Func: Month 12 (n=13,13,9) | 53.49 (8.32) | 47.82 (14.75) | 47.56 (10.97)
  Phys Func: Month 18 (n=15,12,10) | 53.16 (7.68) | 50.29 (11.22) | 44.42 (11.12)
  Phys Func: Month 24 (n=16,13,12) | 50.84 (9.44) | 52.70 (8.47) | 47.39 (9.28)
  Physical: Month 12 (n=13,13,9) | 49.65 (11.30) | 51.85 (10.67) | 42.57 (13.20)
  Physical: Month 18 (n=15,12,10) | 52.01 (8.19) | 50.26 (8.89) | 46.12 (11.37)
  Physical: Month 24 (n=16,13,12) | 48.12 (14.60) | 53.69 (6.69) | 51.45 (6.42)
  Bodily Pain: Month 12 (n=13,13,9) | 53.19 (13.05) | 54.25 (7.34) | 50.70 (11.18)
  Bodily Pain: Month 18 (n=15,12,10) | 53.53 (9.59) | 54.32 (11.78) | 52.64 (10.01)
  Bodily Pain: Month 24 (n=16,13,12) | 53.02 (9.20) | 50.57 (12.55) | 51.51 (8.78)
  General Health: Month 12 (n=12,13,9) | 57.18 (6.12) | 52.96 (8.50) | 47.86 (8.52)
  General Health: Month 18 (n=15,12,10) | 52.54 (10.64) | 50.10 (8.89) | 46.67 (10.08)
  General Health: Month 24 (n=16,13,12) | 49.54 (10.37) | 54.33 (8.23) | 48.14 (6.20)
  Vitality: Month 12 (n=13,13,9) | 59.78 (5.67) | 55.64 (13.28) | 58.61 (11.86)
  Vitality: Month 18 (n=15,12,10) | 53.55 (10.11) | 57.44 (11.69) | 53.75 (10.58)
  Vitality: Month 24 (n=16,13,12) | 54.14 (10.88) | 59.55 (7.19) | 50.96 (9.75)
  Social Function: Month 12 (n=13,13,9) | 48.96 (8.37) | 46.48 (13.14) | 50.43 (9.10)
  Social Function: Month 18 (n=15,12,10) | 49.59 (9.85) | 50.58 (10.11) | 50.49 (12.53)
  Social Function: Month 24 (n=16,13,12) | 51.36 (7.72) | 52.27 (7.00) | 51.03 (9.17)
  Emotional: Month 12 (n=13,13,9) | 49.27 (13.51) | 49.56 (10.54) | 48.53 (10.61)
  Emotional: Month 18 (n=15,12,10) | 51.64 (8.87) | 50.63 (10.12) | 48.49 (12.42)
  Emotional: Month 24 (n=16,13,12) | 47.63 (14.49) | 52.18 (7.16) | 52.52 (4.52)
  Mental Health: Month 12 (n=13,13,9) | 54.05 (8.04) | 51.71 (9.67) | 52.35 (9.08)
  Mental Health: Month 18 (n=15,12,10) | 49.21 (11.37) | 54.66 (9.87) | 49.02 (11.37)
  Mental Health: Month 24 (n=16,13,12) | 51.31 (8.58) | 56.19 (6.45) | 50.50 (9.84)
  TR Scale Score: Month 12 (n=13,13,9) | 1.23 (0.83) | 1.23 (0.83) | 1.33 (1.00)
  TR Scale Score: Month 18 (n=15,12,10) | 1.53 (0.74) | 1.67 (0.78) | 1.70 (1.06)
  TR Scale Score: Month 24 (n=16,13,12) | 2.00 (0.97) | 1.62 (0.77) | 2.33 (0.98)

49. Secondary Outcome: Change From Baseline in SF-36 v2 Subscale Scores by Visit
Description: as for outcome 47
Time Frame: Baseline, Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety Population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 13 | 12 | 10
scores on a scale
  Phys Func: Month 12 (n=13,12,9) | 8.82 (10.58) | 0.51 (12.47) | 5.23 (14.94)
  Phys Func: Month 18 (n=13,10,8) | 9.90 (10.46) | 4.50 (9.92) | 2.56 (15.58)
  Phys Func: Month 24 (n=13,11,10) | 8.48 (10.27) | 3.91 (7.12) | 4.30 (9.86)
  Physical: Month 12 (n=13,12,9) | 13.77 (8.16) | 12.92 (14.51) | 11.67 (14.14)
  Physical: Month 18 (n=13,10,8) | 15.60 (6.36) | 9.54 (9.68) | 12.53 (9.44)
  Physical: Month 24 (n=13,11,10) | 12.30 (8.76) | 13.23 (13.13) | 17.18 (13.81)
  Bodily Pain: Month 12 (n=13,12,9) | 1.47 (15.91) | 6.87 (10.52) | -0.83 (14.54)
  Bodily Pain: Month 18 (n=13,10,8) | 0.83 (11.32) | 8.08 (12.98) | -0.31 (14.06)
  Bodily Pain: Month 24 (n=13,11,10) | 2.56 (10.01) | 5.57 (12.58) | -1.25 (12.99)
  General Health: Month 12 (n=12,11,9) | 11.73 (5.80) | 6.75 (12.04) | 3.60 (7.67)
  General Health: Month 18 (n=13,9,8) | 8.89 (9.64) | 6.94 (8.80) | -1.29 (11.83)
  General Health: Month 24 (n=13,10,10) | 8.06 (8.96) | 9.11 (7.86) | 1.83 (8.55)
  Vitality: Month 12 (n=13,12,9) | 11.05 (9.58) | 9.23 (15.29) | 16.30 (8.87)
  Vitality: Month 18 (n=13,10,8) | 7.14 (13.36) | 11.67 (13.49) | 10.85 (6.96)
  Vitality: Month 24 (n=13,11,8) | 8.90 (10.52) | 15.51 (11.96) | 7.18 (14.06)
  Social Function: Month 12 (n=13,12,9) | 4.14 (10.79) | 7.62 (14.76) | 11.95 (12.55)
  Social Function: Month 18 (n=13,10,8) | 4.55 (14.54) | 11.83 (11.84) | 8.74 (13.77)
  Social Function: Month 24 (n=13,11,10) | 7.03 (12.68) | 11.73 (11.49) | 9.68 (15.38)
  Emotional: Month 12 (n=13,12,9) | 10.19 (13.06) | 7.26 (19.87) | 15.14 (17.45)
  Emotional: Month 18 (n=13,10,8) | 9.32 (15.35) | 11.74 (17.25) | 13.25 (16.56)
  Emotional: Month 24 (n=13,11,10) | 4.66 (17.15) | 6.54 (15.25) | 16.66 (18.82)
  Mental Health: Month 12 (n=13,12,9) | 2.98 (6.64) | 4.62 (8.71) | 5.54 (13.64)
  Mental Health: Month 18 (n=13,10,8) | -1.28 (13.51) | 8.03 (5.76) | 0.00 (14.36)
  Mental Health: Month 24 (n=13,11,10) | 1.70 (9.36) | 10.58 (10.20) | 2.22 (12.72)
  TR Scale Score: Month 12 (n=13,12,9) | -1.31 (1.55) | -1.83 (1.40) | -1.78 (2.11)
  TR Scale Score: Month 18 (n=13,10,8) | -1.15 (1.28) | -1.10 (1.37) | -1.13 (1.81)
  TR Scale Score: Month 24 (n=13,11,10) | -0.92 (1.19) | -1.45 (1.21) | -0.70 (1.25)

50. Secondary Outcome: End Stage Renal Disease Symptom Checklist (ESRD-SCL) Transplanation Module Scores by Visit and Scale
Description: ESRD-SCL: 43-item, disease-specific, self-administered questionnaire. Participants' rated question "At the moment, how much do you suffer?" for each item on 5-point scale, ranged from 0 (not at all) to 4 (extremely). Consisted of 6 subscales: cardiac and renal dysfunction (Range, 0-28), increased growth of gum and hair (Range, 0-20), limited cognitive capacity (Range, 0-32), limited physical capacity (Range, 0-40), side effects (SEs) of corticosteroids (Range, 0-20), transplantation associated psychological distress (TAPD; Range, 0-32); higher scores=greater dysfunction for each subscale. Total score: 0-172, higher scores=greater dysfunction.
Time Frame: Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety Population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 16 | 13 | 11
scores on a scale
  Limited Physical: Month 12 (n = 13, 12, 8) | 0.22 (0.25) | 0.37 (0.40) | 0.29 (0.40)
  Limited Physical: Month 18 (n = 15, 12, 10) | 0.53 (0.69) | 0.41 (0.38) | 0.46 (0.55)
  Limited Physical: Month 24 (n = 16, 13, 11) | 0.60 (0.69) | 0.44 (0.46) | 0.55 (0.46)
  Limited Cognitive: Month 12 (n = 13, 12, 8) | 0.41 (0.40) | 0.45 (0.45) | 0.30 (0.36)
  Limited Cognitive: Month 18 (n = 15, 12, 10) | 0.63 (0.89) | 0.42 (0.42) | 0.29 (0.43)
  Limited Cognitive: Month 24 (n = 16, 13, 11) | 0.65 (0.85) | 0.57 (0.67) | 0.48 (0.54)
  Cardiac / Renal Dysfunc: Month 12 (n = 13, 13, 8) | 0.18 (0.26) | 0.27 (0.31) | 0.18 (0.18)
  Cardiac / Renal Dysfunc: Month 18 (n = 14, 12, 9) | 0.25 (0.38) | 0.30 (0.31) | 0.22 (0.20)
  Cardiac / Renal Dysfunc: Month 24 (n = 15, 13, 11) | 0.33 (0.51) | 0.31 (0.35) | 0.34 (0.24)
  Side effects Corticosteroids: Month 12 (n=13,13,8) | 0.29 (0.35) | 0.57 (0.80) | 0.70 (0.83)
  Side effects Corticosteroids: Month18 (n=14,12,10) | 0.39 (0.65) | 0.45 (0.66) | 0.58 (0.61)
  Side effects Corticosteroids: Month24 (n=15,13,11) | 0.53 (0.64) | 0.26 (0.35) | 0.69 (0.66)
  Increased growth gum/hair: Month 12 (n=13,13,4) | 0.17 (0.24) | 0.15 (0.25) | 0.08 (0.15)
  Increased growth gum/hair: Month 18 (n=15,12,10) | 0.17 (0.28) | 0.23 (0.31) | 0.14 (0.16)
  Increased growth gum/hair: Month 24 (n=16,13,11) | 0.41 (0.49) | 0.28 (0.48) | 0.11 (0.21)
  Transplant-assoc psycho distress:Mnth12(n=13,12,8) | 0.40 (0.42) | 0.50 (0.41) | 0.48 (0.33)
  Transplant-assoc psychodistress:Mnth18(n=15,12,10) | 0.70 (0.81) | 0.42 (0.37) | 0.47 (0.19)
  Transplant-assoc psychodistress:Mnth24(n=16,13,11) | 0.77 (0.72) | 0.45 (0.40) | 0.57 (0.74)
  Global Score: Month 12 (n = 13, 12, 8) | 0.28 (0.26) | 0.39 (0.36) | 0.33 (0.25)
  Global Score: Month 18 (n = 15, 12, 10) | 0.50 (0.65) | 0.38 (0.34) | 0.36 (0.25)
  Global Score: Month 24 (n = 16, 13, 11) | 0.57 (0.59) | 0.40 (0.40) | 0.47 (0.41)

51. Secondary Outcome: Change From Baseline in ESRD-SCL Transplantation Module Scores by Visit and Scale
Description: ESRD-SCL: 43-item, disease-specific, self-administered questionnaire. Participants' rated question "At the moment, how much do you suffer?" for each item on 5-point scale, ranged from 0 (not at all) to 4 (extremely). Consisted of 6 subscales: cardiac and renal dysfunction (Range, 0-28), increased growth of gum and hair (Range, 0-20), limited cognitive capacity (Range, 0-32), limited physical capacity (Range, 0-40), SEs of corticosteroids (Range, 0-20),TAPD (Range, 0-32); higher scores=greater dysfunction for each subscale. Total score: 0-172, higher scores=greater dysfunction.
Time Frame: Baseline, Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety Population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 13 | 10 | 9
scores on a scale
  Limited Physical: Month 12 (n = 13, 10, 8) | -0.34 (0.45) | -0.34 (0.25) | -0.53 (0.38)
  Limited Physical: Month 18 (n = 13, 9, 8) | -0.20 (0.54) | -0.36 (0.32) | -0.30 (0.63)
  Limited Physical: Month 24 (n = 13, 10, 9) | -0.16 (0.63) | -0.23 (0.28) | -0.32 (0.39)
  Limited Cognitive: Month 12 (n = 13, 10, 8) | -0.37 (0.59) | -0.37 (0.24) | -0.36 (0.65)
  Limited Cognitive: Month 18 (n = 13, 9, 8) | -0.22 (0.80) | -0.39 (0.45) | -0.39 (0.54)
  Limited Cognitive: Month 24 (n = 13, 10, 9) | -0.25 (0.89) | -0.21 (0.56) | -0.26 (0.72)
  Cardiac / Renal Dysfunc: Month 12 (n = 13, 9, 8) | -0.48 (0.68) | -0.51 (0.43) | -0.52 (0.49)
  Cardiac / Renal Dysfunc: Month 18 (n = 12, 8, 7) | -0.49 (0.78) | -0.50 (0.41) | -0.45 (0.60)
  Cardiac / Renal Dysfunc: Month 24 (n = 13, 9, 9) | -0.46 (0.61) | -0.41 (0.39) | -0.33 (0.44)
  Side effects Corticosteroids: Month 12(n=13, 9, 8) | -0.25 (0.55) | -0.02 (0.66) | 0.18 (0.61)
  Side effects Corticosteroids: Month 18 (n=12,8,8) | -0.40 (0.72) | -0.23 (0.43) | 0.03 (0.52)
  Side effects Corticosteroids: Month 24 (n=13,10,9) | -0.25 (0.68) | -0.31 (0.55) | 0.13 (0.53)
  Increased growth gum/hair: Month 12 (n=13,10,8) | 0.06 (0.28) | -0.06 (0.40) | -0.08 (0.24)
  Increased growth gum/hair: Month 18 (n=13,9,8) | 0.04 (0.27) | -0.04 (0.46) | -0.03 (0.23)
  Increased growth gum/hair: Month 24 (n=13,10,9) | 0.29 (0.59) | 0.10 (0.63) | -0.07 (0.17)
  Transplant-assoc psychodistress: Mnth12(n=13,10,8) | -0.49 (0.56) | -0.57 (0.58) | -0.61 (0.42)
  Transplant-assoc psychodistress: Mnth18(n=13,9,8) | -0.28 (0.46) | -0.57 (0.55) | -0.48 (0.58)
  Transplant-assoc psychodistress: Mnth24(n=13,10,9) | -0.30 (0.51) | -0.62 (0.67) | -0.61 (0.70)
  Global Score: Month 12 (n = 13, 10, 8) | -0.34 (0.37) | -0.36 (0.24) | -0.37 (0.29)
  Global Score: Month 18 (n = 13, 9, 8) | -0.21 (0.57) | -0.40 (0.31) | -0.31 (0.36)
  Global Score: Month 24 (n = 13, 10, 9) | -0.21 (0.52) | -0.30 (0.31) | -0.28 (0.35)

52. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using Health Care Resource Utilization (HCRU) Questionnaire
Description: HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any number of events including visits to doctor or other healthcare professionals (HCP), non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Months 12, 18, and 24
Population: Safety population; n=number of participants in Safety Population per visit with non-missing value.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Number analyzed (Participants) | 12 | 11 | 9
events
  Doctor/HCP Visits: Month 12 (n=9,10,4) | 3.1 (3.1) | 2.7 (2.5) | 6.3 (3.9)
  Doctor/HCP Visits: Month 18 (n=10,9,6) | 7.2 (9.0) | 6.4 (7.5) | 5.8 (2.7)
  Doctor/HCP Visits: Month 24 (n=12,11,9) | 5.1 (4.2) | 2.5 (2.0) | 5.0 (6.3)
  Other Test/Procedures: Month 12 (n=1,4,4) | 1.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint. | 2.0 (1.4) | 2.3 (1.9)
  Other Test/Procedures: Month 18 (n=4,3,0) | 2.5 (1.7) | 2.0 (1.7) | NA (NA) — No participants were analyzed for this parameter in this treatment group at this timepoint.
  Other Test/Procedures: Month 24 (n=4,3,4) | 3.8 (2.8) | 1.3 (0.6) | 2.8 (2.2)
  Previous Hospitalizations: Month 12 (n=1,1,2) | 2.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint. | 1.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint. | 1.0 (0.0)
  Previous Hospitalizations: Month 18 (n=3,1,1) | 1.3 (0.6) | 1.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint. | 2.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint.
  Previous Hospitalizations: Month 24 (n=3,3,1) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint.
  Emergency Room Visits: Month 12 (n=1,1,2) | 1.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint. | 1.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint. | 1.0 (0.0)
  Emergency Room Visits: Month 18 (n=3,3,1) | 1.3 (0.6) | 1.0 (0.0) | 2.0 (NA) — Measure of dispersion could not be calculated as only 1 participant was analyzed at this timepoint.
  Emergency Room Visits: Month 24 (n=4,2,2) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs; serious and nonserious) were recorded from the time the participant had taken at least 1 dose of trial treatment through the follow-up visit at Month 98 or 2 months following discontinuation of treatment.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tacrolimus | Tofacitinib 15-10-5 mg BID | Tofacitinib 30-15-10 mg BID
Serious Adverse Events (participants affected / at risk) | 7/18 | 10/14 | 8/13
Other Adverse Events (participants affected / at risk) | 17/18 | 14/14 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=18) | Tofacitinib 15-10-5 mg BID (N=14) | Tofacitinib 30-15-10 mg BID (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Transplant rejection (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=18) | Tofacitinib 15-10-5 mg BID (N=14) | Tofacitinib 30-15-10 mg BID (N=13)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 4 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0
Hyphaema (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Asthenia (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 4
Gravitational oedema (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 2
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 5 | 3
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 2
Sluggishness (General disorders) | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
BK virus infection (Infections and infestations) | 1 | 2 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2
Bronchitis viral (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 1
Ear infection (Infections and infestations) | 1 | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 5 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0
Incision site abscess (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 3 | 0
Papilloma viral infection (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 1
Skin candida (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 5
Urinary tract infection (Infections and infestations) | 3 | 5 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Chloracne (Injury, poisoning and procedural complications) | 0 | 0 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2
Arterial bruit (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 1
Blood culture positive (Investigations) | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Cardiac murmur (Investigations) | 0 | 2 | 0
Culture urine positive (Investigations) | 0 | 0 | 1
Electrocardiogram P wave abnormal (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 2
Liver function test abnormal (Investigations) | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
QRS axis abnormal (Investigations) | 1 | 1 | 0
Viral test positive (Investigations) | 1 | 1 | 1
Vitamin D decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 3 | 0
Weight increased (Investigations) | 2 | 1 | 4
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Bone metabolism disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Bowenâ€™s disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Tarsal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 4 | 3
Insomnia (Psychiatric disorders) | 2 | 3 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Kidney fibrosis (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2
Renal cyst (Renal and urinary disorders) | 1 | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0
Renal hypertrophy (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Nipple exudate bloody (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Itching scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Raynaudâ€™s phenomenon (Vascular disorders) | 0 | 1 | 0
Thrombosed varicose vein (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.